CLINICAL TRIAL: NCT02534935
Title: A PHASE 2, RANDOMIZED, CONTROLLED, OBSERVER-BLINDED STUDY CONDUCTED TO DESCRIBE THE IMMUNOGENICITY, SAFETY, AND TOLERABILITY OF A NEISSERIA MENINGITIDIS SEROGROUP B BIVALENT RECOMBINANT LIPOPROTEIN 2086 VACCINE (BIVALENT RLP2086) WHEN ADMINISTERED TO HEALTHY TODDLERS AGED 12 TO <18 MONTHS OR 18 TO <24 MONTHS, AND THE SAFETY AND IMMUNOGENICITY OF A BOOSTER DOSE OF BIVALENT RLP2086
Brief Title: Immunogenicity, Safety and Tolerability of a Neisseria Meningitidis Serogroup B Bivalent Recominant Lipoprotein 2086 Vaccine (Bivalent rLP2086) in Healthy Toddlers.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: B1971035; 2011-004400-38 (EudraCT Number)
Record Dates: First submitted 2015-02-23; First posted 2015-08-28 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-08

CONDITIONS: Meningococcal B Disease
Keywords: Phase 2 Immunogenicity; Safety; Tolerability Study; rLP2086 Vaccine; Healthy Toddlers; Neisseria meningitidis; Duration of Immunogenicity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rLP2086 vaccine (Experimental): Arm stratified by age:
  ≥12 to <18 months and ≥18 to <24 months
  Interventions: Biological: rLP2086 vaccine
- Control (Active Comparator): Arm stratified by age:
  ≥12 to <18 months and ≥18 to <24 months
  Interventions: Biological: Pediatric HAV vaccine

INTERVENTIONS:
Biological: rLP2086 vaccine — 60 mcg or 120mcg at 0, 2 and 6 months
  Arms: rLP2086 vaccine
Biological: Pediatric HAV vaccine — 0.5-mL dose at months 0 and 6. Normal saline at month 2.
  Arms: Control

SUMMARY:
The purpose of this study is to investigate the immunogenicity, safety and tolerability of a new vaccine that might prevent meningococcal B disease. The study will be conducted in healthy toddlers aged between 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged 12 to <15 months or 18 to <24 months during sentinel-cohort enrollment, Or,12 to <24 months during expanded-cohort enrollment.
* Subjects must have received all vaccinations in the relevant National Immunization Program (NIP) for their age group.
* Subject is determined to be in good health by medical history, physical examination, and judgment of the investigator.

Exclusion Criteria:

* Previous vaccination with any meningococcal serogroup B vaccine.
* Previous vaccination with HAV vaccine, or requirement to receive nonstudy HAV vaccine during Stage 1 of the study.
* Contraindication to vaccination with any HAV vaccine or known latex allergy.
* A previous anaphylactic reaction to any vaccine or vaccine-related component.
* Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate intramuscular injection.
* A known or suspected disorder of the immune system that would prevent an immune response to the vaccine, such as subjects with congenital or acquired defects in B-cell function or those receiving systemic immunosuppressive therapy. Subjects with terminal complement deficiency may be included.
* History of microbiologically proven disease caused by N meningitidis or Neisseria gonorrhoeae.
* Significant neurologic disorder or history of seizure (excluding simple febrile seizure).
* Receipt of any blood products, including immunoglobulin, within 6 months before the first study vaccination until the end of Stage 1.
* Current chronic use of systemic antibiotics.
* Received any investigational drugs, vaccines or devices within 28 days before administration of the first study vaccination and/or during study participation.
* Any neuroinflammatory or autoimmune condition, including but not limited to transverse myelitis, uveitis, optic neuritis, and multiple sclerosis.

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 396 (Actual)
Dates: Start 2015-08-31 (Actual); Primary Completion 2017-08-21 (Actual); Study Completion 2020-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (25):
- Australia (6):
  - The Canberra Hospital, Canberra, Garran, Australian Capital Territory
  - Australian Clinical Research Network (ACRN), Maroubra, New South Wales
  - Maroubra Medical Centre, Maroubra, New South Wales
  - Women's And Children's Hospital, North Adelaide, South Australia
  - Murdoch Children's Research Institute, Parkville, Victoria
  - Vaccine Trials Group, Telethon Kids Institute, Perth Children's Hospital, Nedlands, Western Australia
- Czechia (4):
  - Ordinace praktickeho lekare pro deti a dorost, Jindřichův Hradec
  - Samostatna ordinace praktickeho lekare pro deti a dorost, Jindřichův Hradec
  - Medicentrum 6 s.r.o, Praha 6 - Vokovice
  - Prakticky Lekar Pro Deti A Mladez, Týnec nad Sázavou
- Finland (7):
  - Espoo Vaccine Research Clinic, Espoo
  - Helsinki South Vaccine Research Clinic, Helsinki
  - Helsinki East Vaccine Research Clinic, Helsinki
  - Jarvenpaa Vaccine Research Center, Jarvenpaa
  - Pori Vaccine Research Clinic, Pori
  - Tampere Vaccine Research Clinic, Tampere
  - Turku Vaccine Research Clinic, Turku
- Poland (8):
  - NZOZ Vitamed, Bydgoszcz
  - Prywatny Gabinet Lekarski dr n. med. Jerzy Brzostek, Dębica
  - Indywidualna Specjalistyczna Praktyka Lekarska Hanna Czajka, Krakow
  - Specjalistyczna Praktyka Lekarska GRAVITA, Lodz
  - NZOZ Praktyka Lekarza Rodzinnego Eskulap sp. z o.o, Lublin
  - Niepubliczny Zaklad Lecznictwa Ambulatoryjnego Michalkowice Jarosz i Partnerzy Spolka Lekarska, Siemianowice Śląskie
  - Szpital im. Sw. Jadwigi Slaskiej w Trzebnicy Oddzial Pediatryczny, Trzebnica
  - Uniwersytecki Szpital Kliniczny im. J. Mikulicza-Radeckiego we Wroclawiu Klinika Pediatrii i Chorob, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Marshall HS, Vesikari T, Richmond PC, Wysocki J, Szenborn L, Beeslaar J, Maguire JD, Balmer P, O'Neill R, Anderson AS, Pregaldien JL, Maansson R, Jiang HQ, Perez JL. Safety and immunogenicity of a primary series and booster dose of the meningococcal serogroup B-factor H binding protein vaccine (MenB-FHbp) in healthy children aged 1-9 years: two phase 2 randomised, controlled, observer-blinded studies. Lancet Infect Dis. 2023 Jan;23(1):103-116. doi: 10.1016/S1473-3099(22)00424-8. Epub 2022 Sep 7. PMID 36087588
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1971035&StudyName=Immunogenicity%2C%20Safety%20and%20Tolerability%20of%20Meningococcal%20B%20Vaccine%20in%20Healthy%20Toddlers.%20

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In Stage 1, participants received 60 or 120 microgram (mcg) of bivalent rLP2086 vaccine or HAV/saline at Month 1, 2 and 6, and then followed up for 24 months. In Stage 2, participants who received bivalent rLP2086 during Stage 1 had a follow up visit at Month 24. Further participants who received 120 mcg bivalent rLP2086 during Stage 1 were eligible for receiving booster vaccination 6 months after Month 24 visit.
Groups:
- Group 1: 60- mcg Bivalent rLP2086 (>=12 Months to <24 Months): Participants from greater than or equal to (>=) 12 months to less than (<) 24 months of age, received intramuscular injection of 60 mcg of bivalent rLP2086 vaccine on months 0 vaccine on a 0, 2, 6 month schedule.
- Group 2: 120-mcg Bivalent rLP2086 (>=12 Months to <24 Months): Participants from >=12 months to <24 months of age, received intramuscular injection of 120 mcg of bivalent rLP2086 vaccine on a 0, 2, 6 month schedule. All participants who received 3 doses of 120 mcg bivalent rLP2086 in Stage 1 and gave consent for booster vaccination, received intramuscular injection of single booster dose of 120 mcg of bivalent rLP2086 after 23 to 24 months of Vaccination 3, in Stage 2. Participants were followed up approximately 6 months after the booster vaccination.
- Group 3: HAV/Saline (>=12 Months to <24 Months): Stage 1: Participants from >=12 months to <24 months of age, received intramuscular injection of saline on 2 month and HAV vaccine on a 0, 6 month schedule.
Period: Stage 1: 24 Months
Arm/Group | Group 1: 60- mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 2: 120-mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <24 Months): Stage 1
Started | 44 | 220 | 132
Completed | 44 | 210 | 127
Not Completed | 0 | 10 | 5
Not completed — Withdrawal by Subject | 0 | 3 | 3
Not completed — No longer willing to participate in study | 0 | 1 | 1
Not completed — No longer meets eligibility criteria | 0 | 3 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Adverse Event | 0 | 2 | 0
Period: Stage 2: 8 Months
Arm/Group | Group 1: 60- mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 2: 120-mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <24 Months): Stage 1
Started | 40 (Participants entered into Stage 2.) | 174 (Participants who received all 3 doses and entered Stage 2.) | 0 (Participants of HAV/Saline were not eligible for Stage 2.)
Completed | 40 | 170 | 0
Not Completed | 0 | 4 | 0
Not completed — Moved away/parents resigned from study | 0 | 4 | 0
Period: Stage 2: Booster Phase (6 Months)
Arm/Group | Group 1: 60- mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 2: 120-mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <24 Months): Stage 1
Started | 0 (Participants were not eligible for Booster vaccination in Stage 2.) | 148 (Participants who received 3 doses of bivalent rLP2086 in Stage 1 and gave consent for booster vaccination.) | 0 (Participants of HAV/Saline were not eligible for Stage 2.)
Completed | 0 | 147 | 0
Not Completed | 0 | 1 | 0
Not completed — Not received booster vaccination | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of the investigational product (rLP2086, HAV vaccine or saline) and had safety data available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: 60- mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 2: 120-mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <24 Months): Stage 1 | Total
Number analyzed (Participants) | 44 | 220 | 132 | 396
Age, Continuous [Mean (Standard Deviation); unit: months] | 16.9 (4.08) | 17.4 (3.54) | 17.3 (3.58) | 17.3 (3.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 114 | 74 | 209
  Male | 23 | 106 | 58 | 187
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 37 | 210 | 127 | 374
  Race: Asian | 5 | 2 | 1 | 8
  Race: Other | 2 | 8 | 4 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic | 0 | 2 | 0 | 2
  Ethnicity: Non-Hispanic | 44 | 218 | 132 | 394

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Serum Bactericidal Assay Using Human Complement (hSBA) Titers >= Lower Limit of Quantitation (LLOQ) for Each of the 4 Primary Neisseria Meningitidis Serogroup B (MnB) Test Strains 1 Month After Vaccination 3
Description: Percentage of participants achieving hSBA titer >= LLOQ were computed along with corresponding 2-sided 95 percent (%) confidence interval (CIs). LLOQ was 1:16 for PMB80 (A22) and 1:8 for PMB2001 (A56), PMB2948 (B24) and PMB2707 (B44).
Time Frame: 1 month after Vaccination 3
Population: All eligible participants randomized to study received,scheduled investigational products, had pre and post vaccination blood drawn with valid and determinate assay results and had no important protocol deviation. Here,overall number of participants analyzed (N) signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Group 1: 60-µg Bivalent rLP2086 (>=12 Months to <18 Months): Participants from >=12 months to <18 months of age, received intramuscular injection of 60 µg of bivalent rLP2086 vaccine on a 0-, 2-, 6- month schedule.
- Group 1: 60-µg Bivalent rLP2086 (>=18 Months to <24 Months): Participants from >=18 months to <24 months of age, received intramuscular injection of 60 µg of bivalent rLP2086 vaccine on a 0-, 2-, 6- month schedule.
- Group 2: 120-µg Bivalent rLP2086 (>=12 Months to <18 Months): Participants from >=12 months to <18 months of age, received intramuscular injection of 120 µg of bivalent rLP2086 vaccine on a 0-, 2-, 6- month schedule.
- Group 2: 120-µg Bivalent rLP2086 (>=18 Months to <24 Months): Participants from >=18 months to <24 months of age, received intramuscular injection of 120 µg of bivalent rLP2086 vaccine on a 0-, 2-, 6- month schedule.
- Group 3: HAV/Saline (>=12 Months to <18 Months): Participants from >=12 months to <18 months of age, received intramuscular injection of saline on 2- month and HAV vaccine on a 0-, 6- month schedule.
- Group 3: HAV/Saline (>=18 Months to <24 Months): Participants from >=18 months to <24 months of age, received intramuscular injection of saline on 2- month and HAV vaccine on a 0-, 6- month schedule.
Arm/Group | Group 1: 60-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 1: 60-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 2: 120-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 2: 120-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <18 Months) | Group 3: HAV/Saline (>=18 Months to <24 Months)
Number analyzed (Participants) | 9 | 11 | 47 | 51 | 31 | 30
percentage of participants
  PMB80 [A22]: number analyzed (Participants) | 9 | 11 | 45 | 51 | 31 | 29
  PMB80 [A22] | 88.9 [51.8 to 99.7] | 90.9 [58.7 to 99.8] | 91.1 [78.8 to 97.5] | 88.2 [76.1 to 95.6] | 3.2 [0.1 to 16.7] | 6.9 [0.8 to 22.8]
  PMB2001 [A56]: number analyzed (Participants) | 9 | 10 | 47 | 48 | 24 | 30
  PMB2001 [A56] | 100.0 [66.4 to 100.0] | 100.0 [69.2 to 100.0] | 100.0 [92.5 to 100.0] | 100.0 [92.6 to 100.0] | 0.0 [0.0 to 14.2] | 3.3 [0.1 to 17.2]
  PMB2948 [B24]: number analyzed (Participants) | 9 | 11 | 45 | 50 | 31 | 29
  PMB2948 [B24] | 88.9 [51.8 to 99.7] | 81.8 [48.2 to 97.7] | 71.1 [55.7 to 83.6] | 72.0 [57.5 to 83.8] | 3.2 [0.1 to 16.7] | 6.9 [0.8 to 22.8]
  PMB2707 [B44]: number analyzed (Participants) | 9 | 10 | 47 | 47 | 24 | 30
  PMB2707 [B44] | 88.9 [51.8 to 99.7] | 90.0 [55.5 to 99.7] | 87.2 [74.3 to 95.2] | 85.1 [71.7 to 93.8] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 11.6]

2. Primary Outcome: Percentage of Participants Reporting Pre-specified Local Reactions Within 7 Days After Vaccination 1
Description: Local reactions included tenderness at injection site, swelling and redness collected by using an electronic diary (e-diary). Tenderness was graded as: mild (hurted if gently touched), moderate (hurted if gently touched with crying) and severe (caused limitation of limb movement). Redness and swelling were graded as: mild (0.5-2.0 centimeter [cm]), moderate (2.5 to 7.0 cm) and severe (>7.0 cm).
Time Frame: within 7 Days after Vaccination 1
Population: Safety population: all participants who received at least 1 dose of an investigational product (rLP2086 or HAV vaccine) and had safety data available.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: 60-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 1: 60-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 1: 60- mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 2: 120-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 2: 120-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 2: 120-mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <18 Months) | Group 3: HAV/Saline (>=18 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <24 Months): Stage 1
Number analyzed (Participants) | 22 | 22 | 44 | 110 | 110 | 220 | 66 | 66 | 132
percentage of participants
  Tenderness at injection site: Any | 68.2 [45.1 to 86.1] | 50.0 [28.2 to 71.8] | 59.1 [43.2 to 73.7] | 50.9 [41.2 to 60.6] | 64.5 [54.9 to 73.4] | 57.7 [50.9 to 64.3] | 15.2 [7.5 to 26.1] | 19.7 [10.9 to 31.3] | 17.4 [11.4 to 25.0]
  Tenderness at injection site: Mild | 45.5 [24.4 to 67.8] | 27.3 [10.7 to 50.2] | 36.4 [22.4 to 52.2] | 27.3 [19.2 to 36.6] | 34.5 [25.7 to 44.2] | 30.9 [24.9 to 37.5] | 12.1 [5.4 to 22.5] | 19.7 [10.9 to 31.3] | 15.9 [10.1 to 23.3]
  Tenderness at injection site: Moderate | 22.7 [7.8 to 45.4] | 18.2 [5.2 to 40.3] | 20.5 [9.8 to 35.3] | 20.9 [13.7 to 29.7] | 24.5 [16.8 to 33.7] | 22.7 [17.4 to 28.8] | 3.0 [0.4 to 10.5] | 0.0 [0.0 to 5.4] | 1.5 [0.2 to 5.4]
  Tenderness at injection site: Severe | 0.0 [0.0 to 15.4] | 4.5 [0.1 to 22.8] | 2.3 [0.1 to 12.0] | 2.7 [0.6 to 7.8] | 5.5 [2.0 to 11.5] | 4.1 [1.9 to 7.6] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 2.8]
  Redness: Any | 68.2 [45.1 to 86.1] | 40.9 [20.7 to 63.6] | 54.5 [38.8 to 69.6] | 50.9 [41.2 to 60.6] | 42.7 [33.3 to 52.5] | 46.8 [40.1 to 53.6] | 13.6 [6.4 to 24.3] | 16.7 [8.6 to 27.9] | 15.2 [9.5 to 22.4]
  Redness: Mild | 40.9 [20.7 to 63.6] | 27.3 [10.7 to 50.2] | 34.1 [20.5 to 49.9] | 35.5 [26.6 to 45.1] | 21.8 [14.5 to 30.7] | 28.6 [22.8 to 35.1] | 13.6 [6.4 to 24.3] | 16.7 [8.6 to 27.9] | 15.2 [9.5 to 22.4]
  Redness: Moderate | 27.3 [10.7 to 50.2] | 13.6 [2.9 to 34.9] | 20.5 [9.8 to 35.3] | 14.5 [8.5 to 22.5] | 19.1 [12.2 to 27.7] | 16.8 [12.1 to 22.4] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 2.8]
  Redness: Severe | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 0.9 [0.0 to 5.0] | 1.8 [0.2 to 6.4] | 1.4 [0.3 to 3.9] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 2.8]
  Swelling: Any | 36.4 [17.2 to 59.3] | 22.7 [7.8 to 45.4] | 29.5 [16.8 to 45.2] | 30.0 [21.6 to 39.5] | 27.3 [19.2 to 36.6] | 28.6 [22.8 to 35.1] | 7.6 [2.5 to 16.8] | 12.1 [5.4 to 22.5] | 9.8 [5.3 to 16.3]
  Swelling: Mild | 22.7 [7.8 to 45.4] | 13.6 [2.9 to 34.9] | 18.2 [8.2 to 32.7] | 15.5 [9.3 to 23.6] | 19.1 [12.2 to 27.7] | 17.3 [12.5 to 22.9] | 7.6 [2.5 to 16.8] | 12.1 [5.4 to 22.5] | 9.8 [5.3 to 16.3]
  Swelling: Moderate | 13.6 [2.9 to 34.9] | 9.1 [1.1 to 29.2] | 11.4 [3.8 to 24.6] | 13.6 [7.8 to 21.5] | 8.2 [3.8 to 15.0] | 10.9 [7.1 to 15.8] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 2.8]
  Swelling: Severe | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 0.9 [0.0 to 5.0] | 0.0 [0.0 to 3.3] | 0.5 [0.0 to 2.5] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 2.8]

3. Primary Outcome: Percentage of Participants Reporting Pre-specified Local Reactions Within 7 Days After Vaccination 2
Description: Local reactions included tenderness at injection site, swelling and redness collected by using an e-diary. Tenderness was graded as: mild (hurted if gently touched), moderate (hurted if gently touched with crying) and severe (caused limitation of limb movement). Redness and swelling were graded as: mild (0.5-2.0 cm), moderate (2.5 to 7.0 cm) and severe (>7.0 cm).
Time Frame: within 7 Days after Vaccination 2
Population: Safety population: all participants who received at least 1 dose of an investigational product (rLP2086 or HAV vaccine) and had safety data available. Here, N signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | Group 1: 60-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 1: 60-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 1: 60- mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 2: 120-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 2: 120-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 2: 120-mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <18 Months) | Group 3: HAV/Saline (>=18 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <24 Months): Stage 1
Number analyzed (Participants) | 22 | 22 | 44 | 105 | 107 | 212 | 63 | 65 | 128
percentage of Participants
  Tenderness at injection site: Any | 45.5 [24.4 to 67.8] | 50.0 [28.2 to 71.8] | 47.7 [32.5 to 63.3] | 45.7 [36.0 to 55.7] | 60.7 [50.8 to 70.0] | 53.3 [46.3 to 60.2] | 14.3 [6.7 to 25.4] | 15.4 [7.6 to 26.5] | 14.8 [9.2 to 22.2]
  Tenderness at injection site: Mild | 31.8 [13.9 to 54.9] | 40.9 [20.7 to 63.6] | 36.4 [22.4 to 52.2] | 31.4 [22.7 to 41.2] | 32.7 [24.0 to 42.5] | 32.1 [25.8 to 38.8] | 12.7 [5.6 to 23.5] | 15.4 [7.6 to 26.5] | 14.1 [8.6 to 21.3]
  Tenderness at injection site: Moderate | 13.6 [2.9 to 34.9] | 9.1 [1.1 to 29.2] | 11.4 [3.8 to 24.6] | 12.4 [6.8 to 20.2] | 24.3 [16.5 to 33.5] | 18.4 [13.4 to 24.3] | 1.6 [0.0 to 8.5] | 0.0 [0.0 to 5.5] | 0.8 [0.0 to 4.3]
  Tenderness at injection site: Severe | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 1.9 [0.2 to 6.7] | 3.7 [1.0 to 9.3] | 2.8 [1.0 to 6.1] | 0.0 [0.0 to 5.7] | 0.0 [0.0 to 5.5] | 0.0 [0.0 to 2.8]
  Redness: Any | 50.0 [28.2 to 71.8] | 31.8 [13.9 to 54.9] | 40.9 [26.3 to 56.8] | 33.3 [24.4 to 43.2] | 38.3 [29.1 to 48.2] | 35.8 [29.4 to 42.7] | 6.3 [1.8 to 15.5] | 9.2 [3.5 to 19.0] | 7.8 [3.8 to 13.9]
  Redness: Mild | 40.9 [20.7 to 63.6] | 27.3 [10.7 to 50.2] | 34.1 [20.5 to 49.9] | 21.9 [14.4 to 31.0] | 23.4 [15.7 to 32.5] | 22.6 [17.2 to 28.9] | 6.3 [1.8 to 15.5] | 9.2 [3.5 to 19.0] | 7.8 [3.8 to 13.9]
  Redness: Moderate | 9.1 [1.1 to 29.2] | 4.5 [0.1 to 22.8] | 6.8 [1.4 to 18.7] | 11.4 [6.0 to 19.1] | 15.0 [8.8 to 23.1] | 13.2 [9.0 to 18.5] | 0.0 [0.0 to 5.7] | 0.0 [0.0 to 5.5] | 0.0 [0.0 to 2.8]
  Redness: Severe | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 3.4] | 0.0 [0.0 to 1.7] | 0.0 [0.0 to 5.7] | 0.0 [0.0 to 5.5] | 0.0 [0.0 to 2.8]
  Swelling: Any | 18.2 [5.2 to 40.3] | 27.3 [10.7 to 50.2] | 22.7 [11.5 to 37.8] | 21.0 [13.6 to 30.0] | 19.6 [12.6 to 28.4] | 20.3 [15.1 to 26.3] | 1.6 [0.0 to 8.5] | 7.7 [2.5 to 17.0] | 4.7 [1.7 to 9.9]
  Swelling: Mild | 18.2 [5.2 to 40.3] | 13.6 [2.9 to 34.9] | 15.9 [6.6 to 30.1] | 14.3 [8.2 to 22.5] | 13.1 [7.3 to 21.0] | 13.7 [9.4 to 19.1] | 1.6 [0.0 to 8.5] | 7.7 [2.5 to 17.0] | 4.7 [1.7 to 9.9]
  Swelling: Moderate | 0.0 [0.0 to 15.4] | 13.6 [2.9 to 34.9] | 6.8 [1.4 to 18.7] | 6.7 [2.7 to 13.3] | 5.6 [2.1 to 11.8] | 6.1 [3.3 to 10.3] | 0.0 [0.0 to 5.7] | 0.0 [0.0 to 5.5] | 0.0 [0.0 to 2.8]
  Swelling: Severe | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 3.5] | 0.9 [0.0 to 5.1] | 0.5 [0.0 to 2.6] | 0.0 [0.0 to 5.7] | 0.0 [0.0 to 5.5] | 0.0 [0.0 to 2.8]

4. Primary Outcome: Percentage of Participants Reporting Pre-specified Local Reactions Within 7 Days After Vaccination 3
Description: as for outcome 3
Time Frame: within 7 Days after Vaccination 3
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | Group 1: 60-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 1: 60-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 1: 60- mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 2: 120-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 2: 120-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 2: 120-mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <18 Months) | Group 3: HAV/Saline (>=18 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <24 Months): Stage 1
Number analyzed (Participants) | 22 | 22 | 44 | 104 | 108 | 212 | 65 | 63 | 128
percentage of Participants
  Tenderness at injection site: Any | 54.5 [32.2 to 75.6] | 59.1 [36.4 to 79.3] | 56.8 [41.0 to 71.7] | 51.9 [41.9 to 61.8] | 62.0 [52.2 to 71.2] | 57.1 [50.1 to 63.8] | 16.9 [8.8 to 28.3] | 14.3 [6.7 to 25.4] | 15.6 [9.8 to 23.1]
  Tenderness at injection site: Mild | 22.7 [7.8 to 45.4] | 40.9 [20.7 to 63.6] | 31.8 [18.6 to 47.6] | 29.8 [21.2 to 39.6] | 34.3 [25.4 to 44.0] | 32.1 [25.8 to 38.8] | 12.3 [5.5 to 22.8] | 12.7 [5.6 to 23.5] | 12.5 [7.3 to 19.5]
  Tenderness at injection site: Moderate | 31.8 [13.9 to 54.9] | 18.2 [5.2 to 40.3] | 25.0 [13.2 to 40.3] | 17.3 [10.6 to 26.0] | 22.2 [14.8 to 31.2] | 19.8 [14.7 to 25.8] | 4.6 [1.0 to 12.9] | 1.6 [0.0 to 8.5] | 3.1 [0.9 to 7.8]
  Tenderness at injection site: Severe | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 4.8 [1.6 to 10.9] | 5.6 [2.1 to 11.7] | 5.2 [2.6 to 9.1] | 0.0 [0.0 to 5.5] | 0.0 [0.0 to 5.7] | 0.0 [0.0 to 2.8]
  Redness: Any | 40.9 [20.7 to 63.6] | 36.4 [17.2 to 59.3] | 38.6 [24.4 to 54.5] | 32.7 [23.8 to 42.6] | 33.3 [24.6 to 43.1] | 33.0 [26.7 to 39.8] | 7.7 [2.5 to 17.0] | 7.9 [2.6 to 17.6] | 7.8 [3.8 to 13.9]
  Redness: Mild | 31.8 [13.9 to 54.9] | 27.3 [10.7 to 50.2] | 29.5 [16.8 to 45.2] | 23.1 [15.4 to 32.4] | 18.5 [11.7 to 27.1] | 20.8 [15.5 to 26.8] | 6.2 [1.7 to 15.0] | 7.9 [2.6 to 17.6] | 7.0 [3.3 to 12.9]
  Redness: Moderate | 9.1 [1.1 to 29.2] | 9.1 [1.1 to 29.2] | 9.1 [2.5 to 21.7] | 8.7 [4.0 to 15.8] | 14.8 [8.7 to 22.9] | 11.8 [7.8 to 16.9] | 1.5 [0.0 to 8.3] | 0.0 [0.0 to 5.7] | 0.8 [0.0 to 4.3]
  Redness: Severe | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 1.0 [0.0 to 5.2] | 0.0 [0.0 to 3.4] | 0.5 [0.0 to 2.6] | 0.0 [0.0 to 5.5] | 0.0 [0.0 to 5.7] | 0.0 [0.0 to 2.8]
  Swelling: Any | 18.2 [5.2 to 40.3] | 27.3 [10.7 to 50.2] | 22.7 [11.5 to 37.8] | 23.1 [15.4 to 32.4] | 22.2 [14.8 to 31.2] | 22.6 [17.2 to 28.9] | 4.6 [1.0 to 12.9] | 6.3 [1.8 to 15.5] | 5.5 [2.2 to 10.9]
  Swelling: Mild | 9.1 [1.1 to 29.2] | 13.6 [2.9 to 34.9] | 11.4 [3.8 to 24.6] | 16.3 [9.8 to 24.9] | 11.1 [5.9 to 18.6] | 13.7 [9.4 to 19.1] | 4.6 [1.0 to 12.9] | 4.8 [1.0 to 13.3] | 4.7 [1.7 to 9.9]
  Swelling: Moderate | 9.1 [1.1 to 29.2] | 13.6 [2.9 to 34.9] | 11.4 [3.8 to 24.6] | 5.8 [2.1 to 12.1] | 11.1 [5.9 to 18.6] | 8.5 [5.1 to 13.1] | 0.0 [0.0 to 5.5] | 1.6 [0.0 to 8.5] | 0.8 [0.0 to 4.3]
  Swelling: Severe | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 1.0 [0.0 to 5.2] | 0.0 [0.0 to 3.4] | 0.5 [0.0 to 2.6] | 0.0 [0.0 to 5.5] | 0.0 [0.0 to 5.7] | 0.0 [0.0 to 2.8]

5. Primary Outcome: Percentage of Participants Reporting Systemic Events and Antipyretic Use Within 7 Days After Vaccination 1
Description: Systemic reactions included fever, irritability, drowsiness, loss of or decreased appetite and were recorded by using an e-diary. Fever was graded as 38.0 to 38.4 degree Celsius (C), 38.5 to 38.9 degree C, 39.0 to 39.4 degree C, >39.5 to 40.0 degree C and >40.0 degree C. Irritability was graded as mild (easily consolable), moderate (requiring increased attention) and severe (inconsolable). Drowsiness was graded as mild (Increased or prolonged sleeping bouts), moderate (slightly subdued interfering with daily activity) and severe (disabling not interested in usual daily activity). Loss of or decreased appetite was graded as mild (decreased interest in eating), moderate (decreased oral intake) and severe (refusal to feed).
Time Frame: within 7 Days after Vaccination 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | Group 1: 60-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 1: 60-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 1: 60- mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 2: 120-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 2: 120-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 2: 120-mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <18 Months) | Group 3: HAV/Saline (>=18 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <24 Months): Stage 1
Number analyzed (Participants) | 22 | 22 | 44 | 110 | 110 | 220 | 66 | 66 | 132
percentage of Participants
  Fever >=38 degrees C | 40.9 [20.7 to 63.6] | 31.8 [13.9 to 54.9] | 36.4 [22.4 to 52.2] | 28.2 [20.0 to 37.6] | 27.3 [19.2 to 36.6] | 27.7 [21.9 to 34.1] | 10.6 [4.4 to 20.6] | 1.5 [0.0 to 8.2] | 6.1 [2.7 to 11.6]
  Fever 38 to <38.5 degrees C | 22.7 [7.8 to 45.4] | 18.2 [5.2 to 40.3] | 20.5 [9.8 to 35.3] | 7.3 [3.2 to 13.8] | 7.3 [3.2 to 13.8] | 7.3 [4.2 to 11.5] | 6.1 [1.7 to 14.8] | 1.5 [0.0 to 8.2] | 3.8 [1.2 to 8.6]
  Fever 38.5 to <39 degrees C | 13.6 [2.9 to 34.9] | 9.1 [1.1 to 29.2] | 11.4 [3.8 to 24.6] | 14.5 [8.5 to 22.5] | 13.6 [7.8 to 21.5] | 14.1 [9.8 to 19.4] | 1.5 [0.0 to 8.2] | 0.0 [0.0 to 5.4] | 0.8 [0.0 to 4.1]
  Fever 39 to <39.5 degrees C | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 4.5 [1.5 to 10.3] | 3.6 [1.0 to 9.0] | 4.1 [1.9 to 7.6] | 3.0 [0.4 to 10.5] | 0.0 [0.0 to 5.4] | 1.5 [0.2 to 5.4]
  Fever 39.5 to <=40 degrees C | 4.5 [0.1 to 22.8] | 4.5 [0.1 to 22.8] | 4.5 [0.6 to 15.5] | 1.8 [0.2 to 6.4] | 1.8 [0.2 to 6.4] | 1.8 [0.5 to 4.6] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 2.8]
  Fever >40 degrees C | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 3.3] | 0.9 [0.0 to 5.0] | 0.5 [0.0 to 2.5] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 2.8]
  Irritability: Any | 63.6 [40.7 to 82.8] | 50.0 [28.2 to 71.8] | 56.8 [41.0 to 71.7] | 71.8 [62.4 to 80.0] | 60.9 [51.1 to 70.1] | 66.4 [59.7 to 72.6] | 40.9 [29.0 to 53.7] | 33.3 [22.2 to 46.0] | 37.1 [28.9 to 46.0]
  Irritability: Mild | 27.3 [10.7 to 50.2] | 9.1 [1.1 to 29.2] | 18.2 [8.2 to 32.7] | 19.1 [12.2 to 27.7] | 16.4 [10.0 to 24.6] | 17.7 [12.9 to 23.4] | 10.6 [4.4 to 20.6] | 13.6 [6.4 to 24.3] | 12.1 [7.1 to 18.9]
  Irritability: Moderate | 31.8 [13.9 to 54.9] | 40.9 [20.7 to 63.6] | 36.4 [22.4 to 52.2] | 46.4 [36.8 to 56.1] | 39.1 [29.9 to 48.9] | 42.7 [36.1 to 49.6] | 30.3 [19.6 to 42.9] | 16.7 [8.6 to 27.9] | 23.5 [16.5 to 31.6]
  Irritability: Severe | 4.5 [0.1 to 22.8] | 0.0 [0.0 to 15.4] | 2.3 [0.1 to 12.0] | 6.4 [2.6 to 12.7] | 5.5 [2.0 to 11.5] | 5.9 [3.2 to 9.9] | 0.0 [0.0 to 5.4] | 3.0 [0.4 to 10.5] | 1.5 [0.2 to 5.4]
  Drowsiness: Any | 45.5 [24.4 to 67.8] | 40.9 [20.7 to 63.6] | 43.2 [28.3 to 59.0] | 45.5 [35.9 to 55.2] | 42.7 [33.3 to 52.5] | 44.1 [37.4 to 50.9] | 25.8 [15.8 to 38.0] | 10.6 [4.4 to 20.6] | 18.2 [12.0 to 25.8]
  Drowsiness: Mild | 36.4 [17.2 to 59.3] | 31.8 [13.9 to 54.9] | 34.1 [20.5 to 49.9] | 28.2 [20.0 to 37.6] | 24.5 [16.8 to 33.7] | 26.4 [20.7 to 32.7] | 16.7 [8.6 to 27.9] | 6.1 [1.7 to 14.8] | 11.4 [6.5 to 18.0]
  Drowsiness: Moderate | 9.1 [1.1 to 29.2] | 9.1 [1.1 to 29.2] | 9.1 [2.5 to 21.7] | 11.8 [6.4 to 19.4] | 15.5 [9.3 to 23.6] | 13.6 [9.4 to 18.9] | 7.6 [2.5 to 16.8] | 4.5 [0.9 to 12.7] | 6.1 [2.7 to 11.6]
  Drowsiness: Severe | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 5.5 [2.0 to 11.5] | 2.7 [0.6 to 7.8] | 4.1 [1.9 to 7.6] | 1.5 [0.0 to 8.2] | 0.0 [0.0 to 15.4] | 0.8 [0.0 to 4.1]
  Loss of or decrease appetite: Any | 36.4 [17.2 to 59.3] | 36.4 [17.2 to 59.3] | 36.4 [22.4 to 52.2] | 44.5 [35.1 to 54.3] | 46.4 [36.8 to 56.1] | 45.5 [38.7 to 52.3] | 34.8 [23.5 to 47.6] | 10.6 [4.4 to 20.6] | 22.7 [15.9 to 30.8]
  Loss of or decrease appetite: Mild | 22.7 [7.8 to 45.4] | 18.2 [5.2 to 40.3] | 20.5 [9.8 to 35.3] | 16.4 [10.0 to 24.6] | 24.5 [16.8 to 33.7] | 20.5 [15.3 to 26.4] | 13.6 [6.4 to 24.3] | 7.6 [2.5 to 16.8] | 10.6 [5.9 to 17.2]
  Loss of or decrease appetite: Moderate | 13.6 [2.9 to 34.9] | 9.1 [1.1 to 29.2] | 11.4 [3.8 to 24.6] | 25.5 [17.6 to 34.6] | 14.5 [8.5 to 22.5] | 20.0 [14.9 to 25.9] | 18.2 [9.8 to 29.6] | 1.5 [0.0 to 8.2] | 9.8 [5.3 to 16.3]
  Loss of or decrease appetite: Severe | 0.0 [0.0 to 15.4] | 9.1 [1.1 to 29.2] | 4.5 [0.6 to 15.5] | 2.7 [0.6 to 7.8] | 7.3 [3.2 to 13.8] | 5.0 [2.5 to 8.8] | 3.0 [0.4 to 10.5] | 1.5 [0.0 to 8.2] | 2.3 [0.5 to 6.5]
  Antipyretic medication use | 45.5 [24.4 to 67.8] | 59.1 [36.4 to 79.3] | 52.3 [36.7 to 67.5] | 52.7 [43.0 to 62.3] | 40.9 [31.6 to 50.7] | 46.8 [40.1 to 53.6] | 24.2 [14.5 to 36.4] | 15.2 [7.5 to 26.1] | 19.7 [13.3 to 27.5]

6. Primary Outcome: Percentage of Participants Reporting Systemic Events and Antipyretic Use Within 7 Days After Vaccination 2
Description: Systemic reactions included fever, irritability, drowsiness, loss of or decreased appetite and were recorded by using an e-diary. Fever was graded as 38.0 to 38.4 degree C, 38.5 to 38.9 degree C, 39.0 to 39.4 degree C, >39.5 to 40.0 degree C and >40.0 degree C. Irritability was graded as mild (easily consolable), moderate (requiring increased attention) and severe (inconsolable). Drowsiness was graded as mild (Increased or prolonged sleeping bouts), moderate (slightly subdued interfering with daily activity) and severe (disabling not interested in usual daily activity). Loss of or decreased appetite was graded as mild (decreased interest in eating), moderate (decreased oral intake) and severe (refusal to feed).
Time Frame: within 7 Days after Vaccination 2
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | Group 1: 60-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 1: 60-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 1: 60- mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 2: 120-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 2: 120-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 2: 120-mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <18 Months) | Group 3: HAV/Saline (>=18 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <24 Months): Stage 1
Number analyzed (Participants) | 22 | 22 | 44 | 105 | 107 | 212 | 63 | 65 | 128
percentage of Participants
  Fever >=38 degrees C | 13.6 [2.9 to 34.9] | 9.1 [1.1 to 29.2] | 11.4 [3.8 to 24.6] | 14.3 [8.2 to 22.5] | 14.0 [8.1 to 22.1] | 14.2 [9.8 to 19.6] | 6.3 [1.8 to 15.5] | 3.1 [0.4 to 10.7] | 4.7 [1.7 to 9.9]
  Fever 38 to <38.5 degrees C | 13.6 [2.9 to 34.9] | 0.0 [0.0 to 15.4] | 6.8 [1.4 to 18.7] | 4.8 [1.6 to 10.8] | 8.4 [3.9 to 15.4] | 6.6 [3.7 to 10.8] | 4.8 [1.0 to 13.3] | 3.1 [0.4 to 10.7] | 3.9 [1.3 to 8.9]
  Fever 38.5 to <39 degrees C | 0.0 [0.0 to 15.4] | 4.5 [0.1 to 22.8] | 2.3 [0.1 to 12.0] | 6.7 [2.7 to 13.3] | 2.8 [0.6 to 8.0] | 4.7 [2.3 to 8.5] | 1.6 [0.0 to 8.5] | 0.0 [0.0 to 5.5] | 0.8 [0.0 to 4.3]
  Fever 39 to <39.5 degrees C | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 1.9 [0.2 to 6.7] | 1.9 [0.2 to 6.6] | 1.9 [0.5 to 4.8] | 0.0 [0.0 to 5.7] | 0.0 [0.0 to 5.5] | 0.0 [0.0 to 2.8]
  Fever 39.5 to <=40 degrees C | 0.0 [0.0 to 15.4] | 4.5 [0.1 to 22.8] | 2.3 [0.1 to 12.0] | 1.0 [0.0 to 5.2] | 0.9 [0.0 to 5.1] | 0.9 [0.1 to 3.4] | 0.0 [0.0 to 5.7] | 0.0 [0.0 to 5.5] | 0.0 [0.0 to 2.8]
  Fever >40 degrees C | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 3.4] | 0.0 [0.0 to 1.7] | 0.0 [0.0 to 5.7] | 0.0 [0.0 to 5.5] | 0.0 [0.0 to 2.8]
  Irritability: Any | 50.0 [28.2 to 71.8] | 40.9 [20.7 to 63.6] | 45.5 [30.4 to 61.2] | 54.3 [44.3 to 64.0] | 55.1 [45.2 to 64.8] | 54.7 [47.8 to 61.5] | 31.7 [20.6 to 44.7] | 18.5 [9.9 to 30.0] | 25.0 [17.8 to 33.4]
  Irritability: Mild | 40.9 [20.7 to 63.6] | 18.2 [5.2 to 40.3] | 29.5 [16.8 to 45.2] | 19.0 [12.0 to 27.9] | 18.7 [11.8 to 27.4] | 18.9 [13.8 to 24.8] | 7.9 [2.6 to 17.6] | 6.2 [1.7 to 15.0] | 7.0 [3.3 to 12.9]
  Irritability: Moderate | 4.5 [0.1 to 22.8] | 22.7 [7.8 to 45.4] | 13.6 [5.2 to 27.4] | 31.4 [22.7 to 41.2] | 34.6 [25.6 to 44.4] | 33.0 [26.7 to 39.8] | 22.2 [12.7 to 34.5] | 9.2 [3.5 to 19.0] | 15.6 [9.8 to 23.1]
  Irritability: Severe | 4.5 [0.1 to 22.8] | 0.0 [0.0 to 15.4] | 2.3 [0.1 to 12.0] | 3.8 [1.0 to 9.5] | 1.9 [0.2 to 6.6] | 2.8 [1.0 to 6.1] | 1.6 [0.0 to 8.5] | 3.1 [0.4 to 10.7] | 2.3 [0.5 to 6.7]
  Drowsiness: Any | 13.6 [2.9 to 34.9] | 18.2 [5.2 to 40.3] | 15.9 [6.6 to 30.1] | 37.1 [27.9 to 47.1] | 24.3 [16.5 to 33.5] | 30.7 [24.5 to 37.3] | 19.0 [10.2 to 30.9] | 4.6 [1.0 to 12.9] | 11.7 [6.7 to 18.6]
  Drowsiness: Mild | 9.1 [1.1 to 29.2] | 18.2 [5.2 to 40.3] | 13.6 [5.2 to 27.4] | 22.9 [15.2 to 32.1] | 14.0 [8.1 to 22.1] | 18.4 [13.4 to 24.3] | 9.5 [3.6 to 19.6] | 4.6 [1.0 to 12.9] | 7.0 [3.3 to 12.9]
  Drowsiness: Moderate | 4.5 [0.1 to 22.8] | 0.0 [0.0 to 15.4] | 2.3 [0.1 to 12.0] | 13.3 [7.5 to 21.4] | 8.4 [3.9 to 15.4] | 10.8 [7.0 to 15.8] | 7.9 [2.6 to 17.6] | 0.0 [0.0 to 5.5] | 3.9 [1.3 to 8.9]
  Drowsiness: Severe | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 1.0 [0.0 to 5.2] | 1.9 [0.2 to 6.6] | 1.4 [0.3 to 4.1] | 1.6 [0.0 to 8.5] | 0.0 [0.0 to 5.5] | 0.8 [0.0 to 4.3]
  Loss of or decreased appetite: Any | 31.8 [13.9 to 54.9] | 18.2 [5.2 to 40.3] | 25.0 [13.2 to 40.3] | 41.0 [31.5 to 51.0] | 31.8 [23.1 to 41.5] | 36.3 [29.8 to 43.2] | 22.2 [12.7 to 34.5] | 13.8 [6.5 to 24.7] | 18.0 [11.7 to 25.7]
  Loss of or decreased appetite: Mild | 27.3 [10.7 to 50.2] | 18.2 [5.2 to 40.3] | 22.7 [11.5 to 37.8] | 19.0 [12.0 to 27.9] | 19.6 [12.6 to 28.4] | 19.3 [14.3 to 25.3] | 11.1 [4.6 to 21.6] | 7.7 [2.5 to 17.0] | 9.4 [4.9 to 15.8]
  Loss of or decreased appetite: Moderate | 4.5 [0.1 to 22.8] | 0.0 [0.0 to 15.4] | 2.3 [0.1 to 12.0] | 17.1 [10.5 to 25.7] | 7.5 [3.3 to 14.2] | 12.3 [8.2 to 17.5] | 9.5 [3.6 to 19.6] | 6.2 [1.7 to 15.0] | 7.8 [3.8 to 13.9]
  Loss of or decreased appetite: Severe | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 4.8 [1.6 to 10.8] | 4.7 [1.5 to 10.6] | 4.7 [2.3 to 8.5] | 1.6 [0.0 to 8.5] | 0.0 [0.0 to 5.5] | 0.8 [0.0 to 4.3]
  Antipyretic medication use | 45.5 [24.4 to 67.8] | 27.3 [10.7 to 50.2] | 36.4 [22.4 to 52.2] | 35.2 [26.2 to 45.2] | 31.8 [23.1 to 41.5] | 33.5 [27.2 to 40.3] | 19.0 [10.2 to 30.9] | 10.8 [4.4 to 20.9] | 14.8 [9.2 to 22.2]

7. Primary Outcome: Percentage of Participants Reporting Systemic Events and Antipyretic Use Within 7 Days After Vaccination 3
Description: as for outcome 6
Time Frame: within 7 Days after Vaccination 3
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | Group 1: 60-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 1: 60-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 1: 60- mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 2: 120-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 2: 120-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 2: 120-mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <18 Months) | Group 3: HAV/Saline (>=18 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <24 Months): Stage 1
Number analyzed (Participants) | 22 | 22 | 44 | 104 | 108 | 212 | 65 | 63 | 128
percentage of Participants
  Fever >=38 degrees C | 4.5 [0.1 to 22.8] | 4.5 [0.1 to 22.8] | 4.5 [0.6 to 15.5] | 10.6 [5.4 to 18.1] | 14.8 [8.7 to 22.9] | 12.7 [8.6 to 18.0] | 4.6 [1.0 to 12.9] | 7.9 [2.6 to 17.6] | 6.3 [2.7 to 11.9]
  Fever 38 to <38.5 degrees C | 4.5 [0.1 to 22.8] | 4.5 [0.1 to 22.8] | 4.5 [0.6 to 15.5] | 6.7 [2.7 to 13.4] | 6.5 [2.6 to 12.9] | 6.6 [3.7 to 10.8] | 3.1 [0.4 to 10.7] | 4.8 [1.0 to 13.3] | 3.9 [1.3 to 8.9]
  Fever 38.5 to <39 degrees C | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 2.9 [0.6 to 8.2] | 1.9 [0.2 to 6.5] | 2.4 [0.8 to 5.4] | 1.5 [0.0 to 8.3] | 1.6 [0.0 to 8.5] | 1.6 [0.2 to 5.5]
  Fever 39 to <39.5 degrees C | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 1.0 [0.0 to 5.2] | 3.7 [1.0 to 9.2] | 2.4 [0.8 to 5.4] | 0.0 [0.0 to 5.5] | 1.6 [0.0 to 8.5] | 0.8 [0.0 to 4.3]
  Fever 39.5 to <=40 degrees C | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 3.5] | 2.8 [0.6 to 7.9] | 1.4 [0.3 to 4.1] | 0.0 [0.0 to 5.5] | 0.0 [0.0 to 5.7] | 0.0 [0.0 to 2.8]
  Fever >40 degrees C | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 3.4] | 0.0 [0.0 to 1.7] | 0.0 [0.0 to 5.5] | 0.0 [0.0 to 5.7] | 0.0 [0.0 to 2.8]
  Irritability: Any | 36.4 [17.2 to 59.3] | 36.4 [17.2 to 59.3] | 36.4 [22.4 to 52.2] | 56.7 [46.7 to 66.4] | 44.4 [34.9 to 54.3] | 50.5 [43.5 to 57.4] | 24.6 [14.8 to 36.9] | 30.2 [19.2 to 43.0] | 27.3 [19.8 to 35.9]
  Irritability: Mild | 22.7 [7.8 to 45.4] | 18.2 [5.2 to 40.3] | 20.5 [9.8 to 35.3] | 27.9 [19.5 to 37.5] | 19.4 [12.5 to 28.2] | 23.6 [18.0 to 29.9] | 9.2 [3.5 to 19.0] | 15.9 [7.9 to 27.3] | 12.5 [7.3 to 19.5]
  Irritability: Moderate | 13.6 [2.9 to 34.9] | 18.2 [5.2 to 40.3] | 15.9 [6.6 to 30.1] | 26.0 [17.9 to 35.5] | 24.1 [16.4 to 33.3] | 25.0 [19.3 to 31.4] | 13.8 [6.5 to 24.7] | 12.7 [5.6 to 23.5] | 13.3 [7.9 to 20.4]
  Irritability: Severe | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 2.9 [0.6 to 8.2] | 0.9 [0.0 to 5.1] | 1.9 [0.5 to 4.8] | 1.5 [0.0 to 8.3] | 1.6 [0.0 to 8.5] | 1.6 [0.2 to 5.5]
  Drowsiness: Any | 4.5 [0.1 to 22.8] | 22.7 [7.8 to 45.4] | 13.6 [5.2 to 27.4] | 37.5 [28.2 to 47.5] | 30.6 [22.1 to 40.2] | 34.0 [27.6 to 40.8] | 13.8 [6.5 to 24.7] | 12.7 [5.6 to 23.5] | 13.3 [7.9 to 20.4]
  Drowsiness: Mild | 4.5 [0.1 to 22.8] | 22.7 [7.8 to 45.4] | 13.6 [5.2 to 27.4] | 24.0 [16.2 to 33.4] | 23.1 [15.6 to 32.2] | 23.6 [18.0 to 29.9] | 10.8 [4.4 to 20.9] | 9.5 [3.6 to 19.6] | 10.2 [5.5 to 16.7]
  Drowsiness: Moderate | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 10.6 [5.4 to 18.1] | 6.5 [2.6 to 12.9] | 8.5 [5.1 to 13.1] | 3.1 [0.4 to 10.7] | 1.6 [0.0 to 8.5] | 2.3 [0.5 to 6.7]
  Drowsiness: Severe | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 2.9 [0.6 to 8.2] | 0.9 [0.0 to 5.1] | 1.9 [0.5 to 4.8] | 0.0 [0.0 to 5.5] | 1.6 [0.0 to 8.5] | 0.8 [0.0 to 4.3]
  Loss of or decreased appetite: Any | 13.6 [2.9 to 34.9] | 22.7 [7.8 to 45.4] | 18.2 [8.2 to 32.7] | 33.7 [24.7 to 43.6] | 35.2 [26.2 to 45.0] | 34.4 [28.1 to 41.2] | 16.9 [8.8 to 28.3] | 19.0 [10.2 to 30.9] | 18.0 [11.7 to 25.7]
  Loss of or decreased appetite: Mild | 13.6 [2.9 to 34.9] | 22.7 [7.8 to 45.4] | 15.9 [6.6 to 30.1] | 15.4 [9.1 to 23.8] | 18.5 [11.7 to 27.1] | 17.0 [12.2 to 22.7] | 9.2 [3.5 to 19.0] | 15.9 [7.9 to 27.3] | 12.5 [7.3 to 19.5]
  Loss of or decreased appetite: Moderate | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 14.4 [8.3 to 22.7] | 14.8 [8.7 to 22.9] | 14.6 [10.2 to 20.1] | 7.7 [2.5 to 17.0] | 1.6 [0.0 to 8.5] | 4.7 [1.7 to 9.9]
  Loss of or decreased appetite: Severe | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 2.3 [0.1 to 12.0] | 3.8 [1.1 to 9.6] | 1.9 [0.2 to 6.5] | 2.8 [1.0 to 6.1] | 0.0 [0.0 to 5.5] | 1.6 [0.0 to 8.5] | 0.8 [0.0 to 4.3]
  Antipyretic medication use | 18.2 [5.2 to 40.3] | 18.2 [5.2 to 40.3] | 18.2 [8.2 to 32.7] | 34.6 [25.6 to 44.6] | 33.3 [24.6 to 43.1] | 34.0 [27.6 to 40.8] | 13.8 [6.5 to 24.7] | 15.9 [7.9 to 27.3] | 14.8 [9.2 to 22.2]

8. Primary Outcome: Percentage of Participants With at Least 1 Adverse Event (AE), Serious Adverse Event (SAE), Medically Attended Adverse Event (MAE), Newly Diagnosed Chronic Medical Condition (NDCMC) and Immediate Adverse Event (IAE) Within 30 Days After Vaccination 1
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; lack of efficacy in an approved indication; important medical event. A MAE was defined as a non-serious AE that resulted in an evaluation at a medical facility. An NDCMC was defined as a disease or medical condition that was not identified prior to study start and was expected to be persistent or otherwise long-lasting in its effects. Immediate AE was defined as AEs occurring within the first 30 minutes after investigational product administration.
Time Frame: within 30 Days after Vaccination 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | Group 1: 60-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 1: 60-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 1: 60- mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 2: 120-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 2: 120-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 2: 120-mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <18 Months) | Group 3: HAV/Saline (>=18 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <24 Months): Stage 1
Number analyzed (Participants) | 22 | 22 | 44 | 110 | 110 | 220 | 66 | 66 | 132
percentage of Participants
  AE | 18.2 [5.2 to 40.3] | 45.5 [24.4 to 67.8] | 31.8 [18.6 to 47.6] | 38.2 [29.1 to 47.9] | 41.8 [32.5 to 51.6] | 40.0 [33.5 to 46.8] | 33.3 [22.2 to 46.0] | 27.3 [17.0 to 39.6] | 30.3 [22.6 to 38.9]
  SAE | 0.0 [0.0 to 15.4] | 4.5 [0.1 to 22.8] | 2.3 [0.1 to 12.0] | 0.9 [0.0 to 5.0] | 1.8 [0.2 to 6.4] | 1.4 [0.3 to 3.9] | 1.5 [0.0 to 8.2] | 1.5 [0.0 to 8.2] | 1.5 [0.2 to 5.4]
  MAE | 9.1 [1.1 to 29.2] | 13.6 [2.9 to 34.9] | 11.4 [3.8 to 24.6] | 18.2 [11.5 to 26.7] | 19.1 [12.2 to 27.7] | 18.6 [13.7 to 24.4] | 18.2 [9.8 to 29.6] | 16.7 [8.6 to 27.9] | 17.4 [11.4 to 25.0]
  NDCMC | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 3.3] | 0.0 [0.0 to 3.3] | 0.0 [0.0 to 1.7] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 2.8]
  IAE | 0.0 [0.0 to 15.4] | 4.5 [0.1 to 22.8] | 2.3 [0.1 to 12.0] | 0.0 [0.0 to 3.3] | 0.0 [0.0 to 3.3] | 0.0 [0.0 to 1.7] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 2.8]

9. Primary Outcome: Percentage of Participants With at Least 1 Adverse Event (AE), Serious Adverse Event (SAE), Medically Attended Adverse Event (MAE), Newly Diagnosed Chronic Medical Condition (NDCMC) and Immediate Adverse Event (IAE) Within 30 Days After Vaccination 2
Description: as for outcome 8
Time Frame: within 30 Days after Vaccination 2
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | Group 1: 60-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 1: 60-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 1: 60- mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 2: 120-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 2: 120-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 2: 120-mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <18 Months) | Group 3: HAV/Saline (>=18 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <24 Months): Stage 1
Number analyzed (Participants) | 22 | 22 | 44 | 105 | 108 | 213 | 66 | 65 | 131
percentage of Participants
  AE | 18.2 [5.2 to 40.3] | 27.3 [10.7 to 50.2] | 22.7 [11.5 to 37.8] | 34.3 [25.3 to 44.2] | 34.3 [25.4 to 44.0] | 34.3 [27.9 to 41.1] | 24.2 [14.5 to 36.4] | 32.3 [21.2 to 45.1] | 28.2 [20.7 to 36.8]
  SAE | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 3.8 [1.0 to 9.5] | 0.0 [0.0 to 3.4] | 1.9 [0.5 to 4.7] | 1.5 [0.0 to 8.2] | 0.0 [0.0 to 5.5] | 0.8 [0.0 to 4.2]
  MAE | 13.6 [2.9 to 34.9] | 9.1 [1.1 to 29.2] | 11.4 [3.8 to 24.6] | 16.2 [9.7 to 24.7] | 18.5 [11.7 to 27.1] | 17.4 [12.5 to 23.1] | 13.6 [6.4 to 24.3] | 23.1 [13.5 to 35.2] | 18.3 [12.1 to 26.0]
  NDCMC | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 3.4] | 0.0 [0.0 to 1.7] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 5.5] | 0.0 [0.0 to 2.8]
  IAE | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 5.2] | 0.0 [0.0 to 3.4] | 0.5 [0.0 to 2.6] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 5.5] | 0.0 [0.0 to 2.8]

10. Primary Outcome: Percentage of Participants With at Least 1 Adverse Event (AE), Serious Adverse Event (SAE), Medically Attended Adverse Event (MAE), Newly Diagnosed Chronic Medical Condition (NDCMC) and Immediate Adverse Event (IAE) Within 30 Days After Vaccination 3
Description: as for outcome 8
Time Frame: within 30 Days after Vaccination 3
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | Group 1: 60-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 1: 60-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 1: 60- mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 2: 120-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 2: 120-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 2: 120-mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <18 Months) | Group 3: HAV/Saline (>=18 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <24 Months): Stage 1
Number analyzed (Participants) | 22 | 22 | 44 | 104 | 108 | 212 | 65 | 64 | 129
percentage of Participants
  AE | 18.2 [5.2 to 40.3] | 40.9 [20.7 to 63.6] | 29.5 [16.8 to 45.2] | 25.0 [17.0 to 34.4] | 30.6 [22.1 to 40.2] | 27.8 [21.9 to 34.4] | 24.6 [14.8 to 36.9] | 28.1 [17.6 to 40.8] | 26.4 [19.0 to 34.8]
  SAE | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 1.0 [0.0 to 5.2] | 0.0 [0.0 to 3.4] | 0.5 [0.0 to 2.6] | 1.5 [0.0 to 8.3] | 0.0 [0.0 to 5.6] | 0.8 [0.0 to 4.2]
  MAE | 9.1 [1.1 to 29.2] | 27.3 [10.7 to 50.2] | 18.2 [8.2 to 32.7] | 13.5 [7.6 to 21.6] | 16.7 [10.2 to 25.1] | 15.1 [10.6 to 20.6] | 12.3 [5.5 to 22.8] | 20.3 [11.3 to 32.2] | 16.3 [10.4 to 23.8]
  NDCMC | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 3.4] | 0.0 [0.0 to 1.7] | 0.0 [0.0 to 5.5] | 0.0 [0.0 to 5.6] | 0.0 [0.0 to 2.8]
  IAE | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 3.5] | 0.0 [0.0 to 5.1] | 0.5 [0.0 to 2.6] | 0.0 [0.0 to 5.5] | 0.0 [0.0 to 5.6] | 0.0 [0.0 to 2.8]

11. Primary Outcome: Percentage of Participants With at Least 1 Adverse Event (AE), Serious Adverse Event (SAE), Medically Attended Adverse Event (MAE) and Newly Diagnosed Chronic Medical Condition (NDCMC) Within 30 Days After Any Vaccination
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; lack of efficacy in an approved indication; important medical event. A MAE was defined as a non-serious AE that resulted in an evaluation at a medical facility. An NDCMC was defined as a disease or medical condition that was not identified prior to study start and was expected to be persistent or otherwise long-lasting in its effects.
Time Frame: within 30 Days after any Vaccination
Population: Safety population: all participants who received at least 1 dose of the investigational product (rLP2086 or HAV/saline) and had safety data available.
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | Group 1: 60-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 1: 60-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 1: 60- mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 2: 120-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 2: 120-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 2: 120-mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <18 Months) | Group 3: HAV/Saline (>=18 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <24 Months): Stage 1
Number analyzed (Participants) | 22 | 22 | 44 | 110 | 110 | 220 | 66 | 66 | 132
percentage of Participants
  AE | 36.4 [17.2 to 59.3] | 63.6 [40.7 to 82.8] | 50.0 [34.6 to 65.4] | 54.5 [44.8 to 64.1] | 61.8 [52.1 to 70.9] | 58.2 [51.4 to 64.8] | 53.0 [40.3 to 65.4] | 54.5 [41.8 to 66.9] | 53.8 [44.9 to 62.5]
  SAE | 0.0 [0.0 to 15.4] | 4.5 [0.1 to 22.8] | 2.3 [0.1 to 12.0] | 5.5 [2.0 to 11.5] | 1.8 [0.2 to 6.4] | 3.6 [1.6 to 7.0] | 4.5 [0.9 to 12.7] | 1.5 [0.0 to 8.2] | 3.0 [0.8 to 7.6]
  MAE | 22.7 [7.8 to 45.4] | 40.9 [20.7 to 63.6] | 31.8 [18.6 to 47.6] | 32.7 [24.1 to 42.3] | 40.0 [30.8 to 49.8] | 36.4 [30.0 to 43.1] | 31.8 [20.9 to 44.4] | 39.4 [27.6 to 52.2] | 35.6 [27.5 to 44.4]
  NDCMC | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 3.3] | 0.0 [0.0 to 3.3] | 0.0 [0.0 to 1.7] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 2.8]

12. Primary Outcome: Percentage of Participants With at Least 1 Adverse Event (AE), Serious Adverse Event (SAE), Medically Attended Adverse Event (MAE) and Newly Diagnosed Chronic Medical Condition (NDCMC) During the Vaccination Phase
Description: as for outcome 11
Time Frame: From the Vaccination 1 up to 1 month after Vaccination 3
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | Group 1: 60-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 1: 60-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 1: 60- mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 2: 120-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 2: 120-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 2: 120-mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <18 Months) | Group 3: HAV/Saline (>=18 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <24 Months): Stage 1
Number analyzed (Participants) | 22 | 22 | 44 | 110 | 110 | 220 | 66 | 66 | 132
percentage of Participants
  AE | 54.5 [32.2 to 75.6] | 77.3 [54.6 to 92.2] | 65.9 [50.1 to 79.5] | 68.2 [58.6 to 76.7] | 71.8 [62.4 to 80.0] | 70.0 [63.5 to 76.0] | 65.2 [52.4 to 76.5] | 63.6 [50.9 to 75.1] | 64.4 [55.6 to 72.5]
  SAE | 0.0 [0.0 to 15.4] | 9.1 [1.1 to 29.2] | 4.5 [0.6 to 15.5] | 10.9 [5.8 to 18.3] | 3.6 [1.0 to 9.0] | 7.3 [4.2 to 11.5] | 4.5 [0.9 to 12.7] | 6.1 [1.7 to 14.8] | 5.3 [2.2 to 10.6]
  MAE | 36.4 [17.2 to 59.3] | 45.5 [24.4 to 67.8] | 40.9 [26.3 to 56.8] | 47.3 [37.7 to 57.0] | 54.5 [44.8 to 64.1] | 50.9 [44.1 to 57.7] | 42.4 [30.3 to 55.2] | 43.9 [31.7 to 56.7] | 43.2 [34.6 to 52.1]
  NDCMC | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 3.3] | 0.0 [0.0 to 5.0] | 0.5 [0.0 to 2.5] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 2.8]

13. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE), Medically Attended Adverse Event (MAE) and Newly Diagnosed Chronic Medical Condition (NDCMC) During the Follow up Phase
Description: as for outcome 11
Time Frame: From 1 month after Vaccination 3 up to 6 months after Vaccination 3
Population: Safety population: all participants who received at least 1 dose of the investigational product (rLP2086 or HAV/saline) and had safety data available. Here "N" signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | Group 1: 60-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 1: 60-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 1: 60- mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 2: 120-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 2: 120-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 2: 120-mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <18 Months) | Group 3: HAV/Saline (>=18 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <24 Months): Stage 1
Number analyzed (Participants) | 22 | 22 | 44 | 108 | 107 | 215 | 65 | 63 | 128
percentage of Participants
  SAE | 4.5 [0.1 to 22.8] | 9.1 [1.1 to 29.2] | 6.8 [1.4 to 18.7] | 0.9 [0.0 to 5.1] | 3.7 [1.0 to 9.3] | 2.3 [0.8 to 5.3] | 1.5 [0.0 to 8.3] | 1.6 [0.0 to 8.5] | 1.6 [0.2 to 5.5]
  MAE | 22.7 [7.8 to 45.4] | 40.9 [20.7 to 63.6] | 31.8 [18.6 to 47.6] | 29.6 [21.2 to 39.2] | 32.7 [24.0 to 42.5] | 31.2 [25.0 to 37.8] | 30.8 [19.9 to 43.4] | 28.6 [17.9 to 41.3] | 29.7 [21.9 to 38.4]
  NDCMC | 4.5 [0.1 to 22.8] | 0.0 [0.0 to 15.4] | 2.3 [0.1 to 12.0] | 0.0 [0.0 to 3.4] | 0.0 [0.0 to 3.4] | 0.0 [0.0 to 1.7] | 0.0 [0.0 to 5.5] | 0.0 [0.0 to 5.7] | 0.0 [0.0 to 2.8]

14. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE), Medically Attended Adverse Event (MAE) and Newly Diagnosed Chronic Medical Condition (NDCMC) From Vaccination 1 up to 6 Months After Vaccination 3
Description: as for outcome 11
Time Frame: From Vaccination 1 up to 6 months after Vaccination 3
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | Group 1: 60-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 1: 60-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 1: 60- mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 2: 120-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 2: 120-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 2: 120-mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <18 Months) | Group 3: HAV/Saline (>=18 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <24 Months): Stage 1
Number analyzed (Participants) | 22 | 22 | 44 | 110 | 110 | 220 | 66 | 66 | 132
percentage of Participants
  SAE | 4.5 [0.1 to 22.8] | 13.6 [2.9 to 34.9] | 9.1 [2.5 to 21.7] | 10.9 [5.8 to 18.3] | 6.4 [2.6 to 12.7] | 8.6 [5.3 to 13.2] | 6.1 [1.7 to 14.8] | 6.1 [1.7 to 14.8] | 6.1 [2.7 to 11.6]
  MAE | 54.5 [32.2 to 75.6] | 68.2 [45.1 to 86.1] | 61.4 [45.5 to 75.6] | 54.5 [44.8 to 64.1] | 62.7 [53.0 to 71.8] | 58.6 [51.8 to 65.2] | 59.1 [46.3 to 71.0] | 53.0 [40.3 to 65.4] | 56.1 [42.7 to 64.7]
  NDCMC | 4.5 [0.1 to 22.8] | 0.0 [0.0 to 15.4] | 2.3 [0.1 to 12.0] | 0.0 [0.0 to 3.3] | 0.9 [0.0 to 5.0] | 0.5 [0.0 to 2.5] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 2.8]

15. Secondary Outcome: Percentage of Participants With hSBA Titer Between 12 Months to Less Than (<) 24 Months >= LLOQ for Each of the 4 Primary MnB Test Strains at 1, 6, 12, and 24 Months After Vaccination 3
Description: Percentage of participants achieving hSBA titer >= LLOQ were computed along with corresponding 2-sided 95% CIs. LLOQ was 1:16 for PMB80 (A22) and 1:8 for PMB2001 (A56), PMB2948 (B24), and PMB2707 (B44).
Time Frame: 1, 6, 12, 24 months after Vaccination 3
Population: Evaluable immunogenicity population: all eligible participants randomized to study, received scheduled investigational products, had pre and post vaccination blood drawn with valid and determinate assay results and had no important protocol deviation. Here N signifies number of participants evaluable for this outcome measure and "number analyzed" (n) signifies participants evaluable at specific rows.
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | Group 1: 60- mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 2: 120-mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <24 Months): Stage 1
Number analyzed (Participants) | 21 | 97 | 60
percentage of Participants
  PMB80 (A22) 1 Month after Vaccination 3: number analyzed (Participants) | 20 | 96 | 60
  PMB80 (A22) 1 Month after Vaccination 3 | 90.0 [68.3 to 98.8] | 89.6 [81.7 to 94.9] | 5.0 [1.0 to 13.9]
  PMB80 (A22): 6 Months after Vaccination 3: number analyzed (Participants) | 20 | 97 | 58
  PMB80 (A22): 6 Months after Vaccination 3 | 10.0 [1.2 to 31.7] | 12.4 [6.6 to 20.6] | 3.4 [0.4 to 11.9]
  PMB80 (A22): 12 Months after Vaccination 3: number analyzed (Participants) | 21 | 95 | 55
  PMB80 (A22): 12 Months after Vaccination 3 | 14.3 [3.0 to 36.3] | 6.3 [2.4 to 13.2] | 1.8 [0.0 to 9.7]
  PMB80 (A22): 24 Months after Vaccination 3: number analyzed (Participants) | 19 | 81 | 0
  PMB80 (A22): 24 Months after Vaccination 3 | 0.0 [0.0 to 17.6] | 3.7 [0.8 to 10.4] |
  PMB2001 (A56): 1 Month after Vaccination 3: number analyzed (Participants) | 19 | 95 | 54
  PMB2001 (A56): 1 Month after Vaccination 3 | 100.0 [82.4 to 100.0] | 100.0 [96.2 to 100.0] | 1.9 [0.0 to 9.9]
  PMB2001 (A56): 6 months after Vaccination 3: number analyzed (Participants) | 18 | 88 | 52
  PMB2001 (A56): 6 months after Vaccination 3 | 61.1 [35.7 to 82.7] | 59.1 [48.1 to 69.5] | 3.8 [0.5 to 13.2]
  PMB2001 (A56): 12 months after Vaccination 3: number analyzed (Participants) | 16 | 93 | 53
  PMB2001 (A56): 12 months after Vaccination 3 | 56.3 [29.9 to 80.2] | 38.7 [28.8 to 49.4] | 5.7 [1.2 to 15.7]
  PMB2001 (A56): 24 months after Vaccination 3: number analyzed (Participants) | 17 | 79 | 0
  PMB2001 (A56): 24 months after Vaccination 3 | 41.2 [18.4 to 67.1] | 22.8 [14.1 to 33.6] |
  PMB2948 (B24): 1 Month after Vaccination 3: number analyzed (Participants) | 20 | 95 | 60
  PMB2948 (B24): 1 Month after Vaccination 3 | 85.0 [62.1 to 96.8] | 71.6 [61.4 to 80.4] | 5.0 [1.0 to 13.9]
  PMB2948 (B24): 6 month after Vaccination 3: number analyzed (Participants) | 20 | 97 | 58
  PMB2948 (B24): 6 month after Vaccination 3 | 15.0 [3.2 to 37.9] | 10.3 [5.1 to 18.1] | 3.4 [0.4 to 11.9]
  PMB2948 (B24): 12 month after Vaccination 3: number analyzed (Participants) | 21 | 93 | 55
  PMB2948 (B24): 12 month after Vaccination 3 | 9.5 [1.2 to 30.4] | 3.2 [0.7 to 9.1] | 3.6 [0.4 to 12.5]
  PMB2948 (B24): 24 month after Vaccination 3: number analyzed (Participants) | 19 | 82 | 0
  PMB2948 (B24): 24 month after Vaccination 3 | 5.3 [0.1 to 26.0] | 3.7 [0.8 to 10.3] |
  PMB2707 (B44): 1 Month after Vaccination 3: number analyzed (Participants) | 19 | 94 | 54
  PMB2707 (B44): 1 Month after Vaccination 3 | 89.5 [66.9 to 98.7] | 86.2 [77.5 to 92.4] | 0.0 [0.0 to 6.6]
  PMB2707 (B44): 6 month after Vaccination 3: number analyzed (Participants) | 16 | 89 | 53
  PMB2707 (B44): 6 month after Vaccination 3 | 25.0 [7.3 to 52.4] | 40.4 [30.2 to 51.4] | 1.9 [0.0 to 10.1]
  PMB2707 (B44): 12 month after Vaccination 3: number analyzed (Participants) | 16 | 90 | 51
  PMB2707 (B44): 12 month after Vaccination 3 | 12.5 [1.6 to 38.3] | 17.8 [10.5 to 27.3] | 2.0 [0.0 to 10.4]
  PMB2707 (B44): 24 month after Vaccination 3: number analyzed (Participants) | 17 | 80 | 0
  PMB2707 (B44): 24 month after Vaccination 3 | 11.8 [1.5 to 36.4] | 12.5 [6.2 to 21.8] |

16. Secondary Outcome: Percentage of Participants With hSBA Titer >= LLOQ for Each of the 4 Primary MnB Test Strains 1 Month After Vaccination 2
Description: as for outcome 15
Time Frame: 1 month (Mon) after Vaccination (Vac) 2
Population: Evaluable immunogenicity population: all eligible participants randomized to study, received scheduled investigational products, had pre and post vaccination blood drawn with valid and determinate assay results and had no important protocol deviation. Here "N" signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | Group 1: 60-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 1: 60-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 1: 60- mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 2: 120-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 2: 120-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 2: 120-mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <18 Months) | Group 3: HAV/Saline (>=18 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <24 Months): Stage 1
Number analyzed (Participants) | 10 | 10 | 19 | 47 | 50 | 95 | 30 | 29 | 59
percentage of Participants
  1 Mon after Vac2: PMB80[A22]: number analyzed (Participants) | 10 | 9 | 19 | 45 | 50 | 95 | 30 | 29 | 59
  1 Mon after Vac2: PMB80[A22] | 90.0 [55.5 to 99.7] | 66.7 [29.9 to 92.5] | 78.9 [54.4 to 93.9] | 64.4 [48.8 to 78.1] | 84.0 [70.9 to 92.8] | 74.7 [64.8 to 83.1] | 0.0 [0.0 to 11.6] | 3.4 [0.1 to 17.8] | 1.7 [0.0 to 9.1]
  1Mon after Vac2:PMB2001[A56]: number analyzed (Participants) | 9 | 10 | 19 | 47 | 48 | 95 | 23 | 29 | 52
  1Mon after Vac2:PMB2001[A56] | 100.0 [66.4 to 100.0] | 90.0 [55.5 to 99.7] | 94.7 [74.0 to 99.9] | 100.0 [92.5 to 100.0] | 100.0 [92.6 to 100.0] | 100.0 [96.2 to 100.0] | 0.0 [0.0 to 14.8] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 6.8]
  1Mon after Vac2:PMB2948[B24]: number analyzed (Participants) | 10 | 9 | 19 | 42 | 44 | 86 | 30 | 29 | 59
  1Mon after Vac2:PMB2948[B24] | 70.0 [34.8 to 93.3] | 44.4 [13.7 to 78.8] | 57.9 [33.5 to 79.7] | 23.8 [12.1 to 39.5] | 43.2 [28.3 to 59.0] | 33.7 [23.9 to 44.7] | 0.0 [0.0 to 11.6] | 3.4 [0.1 to 17.8] | 1.7 [0.0 to 9.1]
  1Mon after Vac2:PMB2707[B44]: number analyzed (Participants) | 9 | 10 | 19 | 47 | 47 | 94 | 23 | 29 | 52
  1Mon after Vac2:PMB2707[B44] | 77.8 [40.0 to 97.2] | 60.0 [26.2 to 87.8] | 68.4 [43.4 to 87.4] | 72.3 [57.4 to 84.4] | 63.8 [48.5 to 77.3] | 68.1 [57.7 to 77.3] | 0.0 [0.0 to 14.8] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 6.8]

17. Secondary Outcome: Percentage of Participants With Serum Bactericidal Assay Using hSBA Titers >=1:4, >=1:8, >=1:16, >=1:32, >=1:64 and >=1:128 for Each of the 4 Primary Test Strains
Time Frame: Before Vaccination 1 (T1), 1 month after Vaccination 2 (T2), 1 month after Vaccination 3 (T3), 6 months after Vaccination 3 (T4), 12 months after Vaccination 3 (T5) and 24 months after Vaccination 3 (T6)
Population: Evaluable immunogenicity population: all eligible participants randomized to study, received scheduled investigational products, had pre and post vaccination blood drawn with valid and determinate assay results and had no important protocol deviation. Here N signifies number of participants evaluable for this outcome measure and n signifies participants evaluable at specific rows.
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | Group 1: 60-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 1: 60-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 1: 60- mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 2: 120-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 2: 120-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 2: 120-mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <18 Months) | Group 3: HAV/Saline (>=18 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <24 Months): Stage 1
Number analyzed (Participants) | 10 | 11 | 21 | 47 | 51 | 97 | 31 | 30 | 61
percentage of Participants
  T1: PMB80 [A22] - 1:4: number analyzed (Participants) | 9 | 11 | 20 | 46 | 51 | 97 | 31 | 30 | 61
  T1: PMB80 [A22] - 1:4 | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 16.8] | 4.3 [0.5 to 14.8] | 3.9 [0.5 to 13.5] | 4.1 [1.1 to 10.2] | 0.0 [0.0 to 11.2] | 3.3 [0.1 to 17.2] | 1.6 [0.0 to 8.8]
  T1: PMB80 [A22] - 1:8: number analyzed (Participants) | 9 | 11 | 20 | 46 | 51 | 97 | 31 | 30 | 61
  T1: PMB80 [A22] - 1:8 | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 16.8] | 2.2 [0.1 to 11.5] | 3.9 [0.5 to 13.5] | 3.1 [0.6 to 8.8] | 0.0 [0.0 to 11.2] | 3.3 [0.1 to 17.2] | 1.6 [0.0 to 8.8]
  T1: PMB80 [A22] - 1:16: number analyzed (Participants) | 9 | 11 | 20 | 46 | 51 | 97 | 31 | 30 | 61
  T1: PMB80 [A22] - 1:16 | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 16.8] | 2.2 [0.1 to 11.5] | 3.9 [0.5 to 13.5] | 3.1 [0.6 to 8.8] | 0.0 [0.0 to 11.2] | 3.3 [0.1 to 17.2] | 1.6 [0.0 to 8.8]
  T1: PMB80 [A22] - 1:32: number analyzed (Participants) | 9 | 11 | 20 | 46 | 51 | 97 | 31 | 30 | 61
  T1: PMB80 [A22] - 1:32 | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 16.8] | 2.2 [0.1 to 11.5] | 2.0 [0.0 to 10.4] | 2.1 [0.3 to 7.3] | 0.0 [0.0 to 11.2] | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 5.9]
  T1: PMB80 [A22] - 1:64: number analyzed (Participants) | 9 | 11 | 20 | 46 | 51 | 97 | 31 | 30 | 61
  T1: PMB80 [A22] - 1:64 | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 16.8] | 2.2 [0.1 to 11.5] | 0.0 [0.0 to 7.0] | 1.0 [0.0 to 5.6] | 0.0 [0.0 to 11.2] | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 5.9]
  T1: PMB80 [A22] - 1:128: number analyzed (Participants) | 9 | 11 | 20 | 46 | 51 | 97 | 31 | 30 | 61
  T1: PMB80 [A22] - 1:128 | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 16.8] | 2.2 [0.1 to 11.5] | 0.0 [0.0 to 7.0] | 1.0 [0.0 to 5.6] | 0.0 [0.0 to 11.2] | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 5.9]
  T1: PMB2001 (A56)-1:4: number analyzed (Participants) | 9 | 10 | 19 | 46 | 49 | 95 | 24 | 29 | 53
  T1: PMB2001 (A56)-1:4 | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 7.7] | 4.1 [0.5 to 14.0] | 2.1 [0.3 to 7.4] | 4.2 [0.1 to 21.1] | 0.0 [0.0 to 11.9] | 1.9 [0.0 to 10.1]
  T1: PMB2001 (A56)-1:8: number analyzed (Participants) | 9 | 10 | 19 | 46 | 49 | 95 | 24 | 29 | 53
  T1: PMB2001 (A56)-1:8 | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 7.7] | 2.0 [0.1 to 10.9] | 1.1 [0.0 to 5.7] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 6.7]
  T1: PMB2001 (A56)-1:16: number analyzed (Participants) | 9 | 10 | 19 | 46 | 49 | 95 | 24 | 29 | 53
  T1: PMB2001 (A56)-1:16 | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 7.7] | 2.0 [0.1 to 10.9] | 1.1 [0.0 to 5.7] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 6.7]
  T1: PMB2001 (A56)-1:32: number analyzed (Participants) | 9 | 10 | 19 | 46 | 49 | 95 | 24 | 29 | 53
  T1: PMB2001 (A56)-1:32 | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 7.7] | 2.0 [0.1 to 10.9] | 1.1 [0.0 to 5.7] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 6.7]
  T1: PMB2001 (A56)-1:64: number analyzed (Participants) | 9 | 10 | 19 | 46 | 49 | 95 | 24 | 29 | 53
  T1: PMB2001 (A56)-1:64 | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 7.7] | 0.0 [0.0 to 7.3] | 0.0 [0.0 to 3.8] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 6.7]
  T1: PMB2001 (A56)-1:128: number analyzed (Participants) | 9 | 10 | 19 | 46 | 49 | 95 | 24 | 29 | 53
  T1: PMB2001 (A56)-1:128 | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 7.7] | 0.0 [0.0 to 7.3] | 0.0 [0.0 to 3.8] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 6.7]
  T1: PMB2948 (B24)-1:4: number analyzed (Participants) | 10 | 11 | 21 | 46 | 51 | 97 | 31 | 30 | 61
  T1: PMB2948 (B24)-1:4 | 0.0 [0.0 to 30.8] | 9.1 [0.2 to 41.3] | 4.8 [0.1 to 23.8] | 2.2 [0.1 to 11.5] | 2.0 [0.0 to 10.4] | 2.1 [0.3 to 7.3] | 0.0 [0.0 to 11.2] | 3.3 [0.1 to 17.2] | 1.6 [0.0 to 8.8]
  T1: PMB2948 (B24)-1:8: number analyzed (Participants) | 10 | 11 | 21 | 46 | 51 | 97 | 31 | 30 | 61
  T1: PMB2948 (B24)-1:8 | 0.0 [0.0 to 30.8] | 9.1 [0.2 to 41.3] | 4.8 [0.1 to 23.8] | 2.2 [0.1 to 11.5] | 2.0 [0.0 to 10.4] | 2.1 [0.3 to 7.3] | 0.0 [0.0 to 11.2] | 3.3 [0.1 to 17.2] | 1.6 [0.0 to 8.8]
  T1: PMB2948 (B24)-1:16: number analyzed (Participants) | 10 | 11 | 21 | 46 | 51 | 97 | 31 | 30 | 61
  T1: PMB2948 (B24)-1:16 | 0.0 [0.0 to 30.8] | 9.1 [0.2 to 41.3] | 4.8 [0.1 to 23.8] | 2.2 [0.1 to 11.5] | 2.0 [0.0 to 10.4] | 2.1 [0.3 to 7.3] | 0.0 [0.0 to 11.2] | 3.3 [0.1 to 17.2] | 1.6 [0.0 to 8.8]
  T1: PMB2948 (B24)-1:32: number analyzed (Participants) | 10 | 11 | 21 | 46 | 51 | 97 | 31 | 30 | 61
  T1: PMB2948 (B24)-1:32 | 0.0 [0.0 to 30.8] | 9.1 [0.2 to 14.3] | 4.8 [0.1 to 23.8] | 0.0 [0.0 to 7.7] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 3.7] | 0.0 [0.0 to 11.2] | 3.3 [0.1 to 17.2] | 1.6 [0.0 to 8.8]
  T1: PMB2948 (B24)-1:64: number analyzed (Participants) | 10 | 11 | 21 | 46 | 51 | 97 | 31 | 30 | 61
  T1: PMB2948 (B24)-1:64 | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 7.7] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 3.7] | 0.0 [0.0 to 11.2] | 3.3 [0.1 to 17.2] | 1.6 [0.0 to 8.8]
  T1: PMB2948 (B24)-1:128: number analyzed (Participants) | 10 | 11 | 21 | 46 | 51 | 97 | 31 | 30 | 61
  T1: PMB2948 (B24)-1:128 | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 7.7] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 3.7] | 0.0 [0.0 to 11.2] | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 5.9]
  T1: PMB2707 (B44)-1:4: number analyzed (Participants) | 9 | 10 | 19 | 46 | 49 | 95 | 24 | 30 | 54
  T1: PMB2707 (B44)-1:4 | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 17.6] | 2.2 [0.1 to 11.5] | 0.0 [0.0 to 7.3] | 1.1 [0.0 to 5.7] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 6.6]
  T1: PMB2707 (B44)-1:8: number analyzed (Participants) | 9 | 10 | 19 | 46 | 49 | 95 | 24 | 30 | 54
  T1: PMB2707 (B44)-1:8 | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 17.6] | 2.2 [0.1 to 11.5] | 0.0 [0.0 to 7.3] | 1.1 [0.0 to 5.7] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 6.6]
  T1: PMB2707 (B44)-1:16: number analyzed (Participants) | 9 | 10 | 19 | 46 | 49 | 95 | 24 | 30 | 54
  T1: PMB2707 (B44)-1:16 | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 7.7] | 0.0 [0.0 to 7.3] | 0.0 [0.0 to 3.8] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 6.6]
  T1: PMB2707 (B44)-1:32: number analyzed (Participants) | 9 | 10 | 19 | 46 | 49 | 95 | 24 | 30 | 54
  T1: PMB2707 (B44)-1:32 | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 7.7] | 0.0 [0.0 to 7.3] | 0.0 [0.0 to 3.8] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 6.6]
  T1: PMB2707 (B44)-1:64: number analyzed (Participants) | 9 | 10 | 19 | 46 | 49 | 95 | 24 | 30 | 54
  T1: PMB2707 (B44)-1:64 | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 7.7] | 0.0 [0.0 to 7.3] | 0.0 [0.0 to 3.8] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 6.6]
  T1: PMB2707 (B44)-1:128: number analyzed (Participants) | 9 | 10 | 19 | 46 | 49 | 95 | 24 | 30 | 54
  T1: PMB2707 (B44)-1:128 | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 7.7] | 0.0 [0.0 to 7.3] | 0.0 [0.0 to 3.8] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 6.6]
  T2: PMB80 [A22] - 1:4: number analyzed (Participants) | 10 | 9 | 19 | 45 | 50 | 95 | 30 | 29 | 59
  T2: PMB80 [A22] - 1:4 | 90.0 [55.5 to 99.7] | 66.7 [29.9 to 92.5] | 78.9 [54.4 to 93.9] | 64.4 [48.8 to 78.1] | 86.0 [73.3 to 94.2] | 75.8 [65.9 to 84.0] | 0.0 [0.0 to 11.6] | 3.4 [0.1 to 17.8] | 1.7 [0.0 to 9.1]
  T2: PMB80 [A22] - 1:8: number analyzed (Participants) | 10 | 9 | 19 | 45 | 50 | 95 | 30 | 29 | 59
  T2: PMB80 [A22] - 1:8 | 90.0 [55.5 to 99.7] | 66.7 [29.9 to 92.5] | 78.9 [54.4 to 93.9] | 64.4 [48.8 to 78.1] | 86.0 [73.3 to 94.2] | 75.8 [65.9 to 84.0] | 0.0 [0.0 to 11.6] | 3.4 [0.1 to 17.8] | 1.7 [0.0 to 9.1]
  T2: PMB80 [A22] - 1:32: number analyzed (Participants) | 10 | 9 | 19 | 45 | 50 | 95 | 30 | 29 | 59
  T2: PMB80 [A22] - 1:32 | 80.0 [44.4 to 97.5] | 44.4 [13.7 to 78.8] | 63.2 [38.4 to 83.7] | 51.1 [35.8 to 66.3] | 66.0 [51.2 to 78.8] | 58.9 [48.4 to 68.9] | 0.0 [0.0 to 11.6] | 3.4 [0.1 to 17.8] | 1.7 [0.0 to 9.1]
  T2: PMB80 [A22] - 1:64: number analyzed (Participants) | 10 | 9 | 19 | 45 | 50 | 95 | 30 | 29 | 59
  T2: PMB80 [A22] - 1:64 | 50.0 [18.7 to 81.3] | 22.2 [2.8 to 60.0] | 36.8 [16.3 to 61.6] | 28.9 [16.4 to 44.3] | 40.0 [26.4 to 54.8] | 34.7 [25.3 to 45.2] | 0.0 [0.0 to 11.6] | 3.4 [0.1 to 17.8] | 1.7 [0.0 to 9.1]
  T2: PMB80 [A22] - 1:128: number analyzed (Participants) | 10 | 9 | 19 | 45 | 50 | 95 | 30 | 29 | 59
  T2: PMB80 [A22] - 1:128 | 20.0 [2.5 to 55.6] | 22.2 [2.8 to 60.0] | 21.1 [6.1 to 45.6] | 11.1 [3.7 to 24.1] | 16.0 [7.2 to 29.1] | 13.7 [7.5 to 22.3] | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 6.1]
  T2: PMB2001 [A56]- 1:4: number analyzed (Participants) | 9 | 10 | 19 | 47 | 48 | 95 | 23 | 29 | 52
  T2: PMB2001 [A56]- 1:4 | 100.0 [66.4 to 100.0] | 100.0 [69.2 to 100.0] | 100.0 [82.4 to 100.0] | 100.0 [92.5 to 100.0] | 100.0 [92.6 to 100.0] | 100.0 [96.2 to 100.0] | 4.3 [0.1 to 21.9] | 0.0 [0.0 to 11.9] | 1.9 [0.0 to 10.3]
  T2: PMB2001 [A56]- 1:16: number analyzed (Participants) | 9 | 10 | 19 | 47 | 48 | 95 | 23 | 29 | 52
  T2: PMB2001 [A56]- 1:16 | 100.0 [66.4 to 100.0] | 90.0 [55.5 to 99.7] | 94.7 [74.0 to 99.9] | 100.0 [92.5 to 100.0] | 100.0 [92.6 to 100.0] | 100.0 [96.2 to 100.0] | 0.0 [0.0 to 14.8] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 6.8]
  T2: PMB2001 [A56]- 1:32: number analyzed (Participants) | 9 | 10 | 19 | 47 | 48 | 95 | 23 | 29 | 52
  T2: PMB2001 [A56]- 1:32 | 100.0 [66.4 to 100.0] | 90.0 [55.5 to 99.7] | 94.7 [74.0 to 99.9] | 95.7 [85.5 to 99.5] | 95.8 [85.7 to 99.5] | 95.8 [89.6 to 98.8] | 0.0 [0.0 to 14.8] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 6.8]
  T2:PMB2001 [A56]- 1:64: number analyzed (Participants) | 9 | 10 | 19 | 47 | 48 | 95 | 23 | 29 | 52
  T2:PMB2001 [A56]- 1:64 | 100.0 [66.4 to 100.0] | 70.0 [34.8 to 93.3] | 84.2 [60.4 to 96.6] | 87.2 [74.3 to 95.2] | 85.4 [72.2 to 93.9] | 86.3 [77.7 to 92.5] | 0.0 [0.0 to 14.8] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 6.8]
  T2:PMB2001 [A56]-1:128: number analyzed (Participants) | 9 | 10 | 19 | 47 | 48 | 95 | 23 | 29 | 52
  T2:PMB2001 [A56]-1:128 | 44.4 [13.7 to 78.8] | 50.0 [18.7 to 81.3] | 47.4 [24.4 to 71.1] | 59.6 [44.3 to 73.6] | 54.2 [39.2 to 68.8] | 56.8 [46.3 to 67.0] | 0.0 [0.0 to 14.8] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 6.8]
  T2: PMB2948 (B24)-1:4: number analyzed (Participants) | 10 | 9 | 19 | 42 | 44 | 86 | 30 | 29 | 59
  T2: PMB2948 (B24)-1:4 | 70.0 [34.8 to 93.3] | 44.4 [13.7 to 78.8] | 57.9 [33.5 to 79.7] | 28.6 [15.7 to 44.6] | 43.2 [28.3 to 59.0] | 36.0 [26.0 to 47.1] | 0.0 [0.0 to 11.6] | 3.4 [0.1 to 17.8] | 1.7 [0.0 to 9.1]
  T2: PMB2948 (B24)-1:16: number analyzed (Participants) | 10 | 9 | 19 | 42 | 44 | 86 | 30 | 29 | 59
  T2: PMB2948 (B24)-1:16 | 60.0 [26.2 to 87.8] | 33.3 [7.5 to 70.1] | 47.4 [24.4 to 71.7] | 21.4 [10.3 to 36.8] | 43.2 [28.3 to 59.0] | 32.6 [22.8 to 43.5] | 0.0 [0.0 to 11.6] | 3.4 [0.1 to 17.8] | 1.7 [0.0 to 9.1]
  T2: PMB2948 (B24)-1:32: number analyzed (Participants) | 10 | 9 | 19 | 42 | 44 | 86 | 30 | 29 | 59
  T2: PMB2948 (B24)-1:32 | 10.0 [0.3 to 44.5] | 0.0 [0.0 to 33.6] | 5.3 [0.1 to 26.0] | 9.5 [2.7 to 22.6] | 18.2 [8.2 to 32.7] | 14.0 [7.4 to 23.1] | 0.0 [0.0 to 11.6] | 3.4 [0.1 to 17.8] | 1.7 [0.0 to 9.1]
  T2: PMB2948 (B24)-1:64: number analyzed (Participants) | 10 | 9 | 19 | 42 | 44 | 86 | 30 | 29 | 59
  T2: PMB2948 (B24)-1:64 | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 17.6] | 2.4 [0.1 to 12.6] | 4.5 [0.6 to 15.5] | 3.5 [0.7 to 9.9] | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 6.1]
  T2: PMB2948 (B24)-1:128: number analyzed (Participants) | 10 | 9 | 19 | 42 | 44 | 86 | 30 | 29 | 59
  T2: PMB2948 (B24)-1:128 | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 17.6] | 2.4 [0.1 to 12.6] | 0.0 [0.0 to 8.0] | 1.2 [0.0 to 6.3] | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 6.1]
  T2: PMB2707 (B44)-1:4: number analyzed (Participants) | 9 | 10 | 19 | 47 | 47 | 94 | 23 | 29 | 52
  T2: PMB2707 (B44)-1:4 | 77.8 [40.0 to 97.2] | 70.0 [34.8 to 93.3] | 73.7 [48.8 to 90.9] | 72.3 [57.4 to 84.4] | 63.8 [48.5 to 77.3] | 68.1 [57.7 to 77.3] | 0.0 [0.0 to 14.8] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 6.8]
  T2: PMB2707 (B44)-1:16: number analyzed (Participants) | 9 | 10 | 19 | 47 | 47 | 94 | 23 | 29 | 52
  T2: PMB2707 (B44)-1:16 | 77.8 [40.0 to 97.2] | 60.0 [26.2 to 87.8] | 68.4 [43.4 to 87.4] | 72.3 [57.4 to 84.4] | 61.7 [46.4 to 75.5] | 67.0 [56.6 to 76.4] | 0.0 [0.0 to 14.8] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 6.8]
  T2: PMB2707 (B44)-1:32: number analyzed (Participants) | 9 | 10 | 19 | 47 | 47 | 94 | 23 | 29 | 52
  T2: PMB2707 (B44)-1:32 | 55.6 [21.2 to 86.3] | 60.0 [26.2 to 87.8] | 57.9 [33.5 to 79.7] | 61.7 [46.4 to 75.5] | 51.1 [36.1 to 65.9] | 56.4 [45.8 to 66.6] | 0.0 [0.0 to 14.8] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 6.8]
  T2: PMB2707 (B44)-1:64: number analyzed (Participants) | 9 | 10 | 19 | 47 | 47 | 94 | 23 | 29 | 52
  T2: PMB2707 (B44)-1:64 | 33.3 [7.5 to 70.1] | 30.0 [6.7 to 65.2] | 31.6 [12.6 to 56.6] | 27.7 [15.6 to 42.6] | 21.3 [10.7 to 35.7] | 24.5 [16.2 to 34.4] | 0.0 [0.0 to 14.8] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 6.8]
  T2: PMB2707 (B44)-1:128: number analyzed (Participants) | 9 | 10 | 19 | 47 | 47 | 94 | 23 | 29 | 52
  T2: PMB2707 (B44)-1:128 | 11.1 [0.3 to 48.2] | 10.0 [0.3 to 44.5] | 10.5 [1.3 to 33.1] | 10.6 [3.5 to 23.1] | 10.6 [3.5 to 23.1] | 10.6 [5.2 to 18.7] | 0.0 [0.0 to 14.8] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 6.8]
  T3: PMB80 (A22)-1:4: number analyzed (Participants) | 9 | 11 | 20 | 45 | 51 | 96 | 31 | 29 | 60
  T3: PMB80 (A22)-1:4 | 88.9 [51.8 to 99.7] | 90.9 [58.7 to 99.8] | 90.0 [68.3 to 98.8] | 91.1 [78.8 to 97.5] | 88.2 [76.1 to 95.6] | 89.6 [81.7 to 94.9] | 6.5 [0.8 to 21.4] | 6.9 [0.8 to 22.8] | 6.7 [1.8 to 16.2]
  T3: PMB80 (A22)-1:8: number analyzed (Participants) | 9 | 11 | 20 | 45 | 51 | 96 | 31 | 29 | 60
  T3: PMB80 (A22)-1:8 | 88.9 [51.8 to 99.7] | 90.9 [58.7 to 99.8] | 90.0 [68.3 to 98.8] | 91.1 [78.8 to 97.5] | 88.2 [76.1 to 95.6] | 89.6 [81.7 to 94.9] | 6.5 [0.8 to 21.4] | 6.9 [0.8 to 22.8] | 6.7 [1.8 to 16.2]
  T3: PMB80 (A22)-1:32: number analyzed (Participants) | 9 | 11 | 20 | 45 | 51 | 96 | 31 | 29 | 60
  T3: PMB80 (A22)-1:32 | 88.9 [51.8 to 99.7] | 81.8 [48.2 to 97.7] | 85.0 [62.1 to 96.8] | 82.2 [67.9 to 92.0] | 86.3 [73.7 to 94.3] | 84.4 [75.5 to 91.0] | 3.2 [0.1 to 16.7] | 3.4 [0.1 to 17.8] | 3.3 [0.4 to 11.5]
  T3: PMB80 (A22)-1:64: number analyzed (Participants) | 9 | 11 | 20 | 45 | 51 | 96 | 31 | 29 | 60
  T3: PMB80 (A22)-1:64 | 66.7 [29.9 to 92.5] | 72.7 [39.0 to 94.0] | 70.0 [45.7 to 88.1] | 60.0 [44.3 to 74.3] | 72.5 [58.3 to 84.1] | 66.7 [56.3 to 76.0] | 3.2 [0.1 to 16.7] | 0.0 [0.0 to 11.9] | 1.7 [0.0 to 8.9]
  T3: PMB80 (A22)-1:128: number analyzed (Participants) | 9 | 11 | 20 | 45 | 51 | 96 | 31 | 29 | 60
  T3: PMB80 (A22)-1:128 | 44.4 [13.7 to 78.8] | 54.5 [23.4 to 83.3] | 50.0 [27.2 to 72.8] | 37.8 [23.8 to 53.5] | 49.0 [34.8 to 63.4] | 43.8 [33.6 to 54.3] | 0.0 [0.0 to 11.2] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 6.0]
  T3: PMB2001 (A56)-1:4: number analyzed (Participants) | 9 | 10 | 19 | 47 | 48 | 95 | 24 | 30 | 54
  T3: PMB2001 (A56)-1:4 | 100.0 [66.4 to 100.0] | 100.0 [69.2 to 100.0] | 100.0 [82.4 to 100.0] | 100.0 [92.5 to 100.0] | 100.0 [92.6 to 100.0] | 100.0 [96.2 to 100.0] | 8.3 [1.0 to 27.0] | 10.0 [2.1 to 26.5] | 9.3 [3.1 to 20.3]
  T3: PMB2001 (A56)-1:16: number analyzed (Participants) | 9 | 10 | 19 | 47 | 48 | 95 | 24 | 30 | 54
  T3: PMB2001 (A56)-1:16 | 100.0 [66.4 to 100.0] | 100.0 [69.2 to 100.0] | 100.0 [82.4 to 100.0] | 97.9 [88.7 to 99.9] | 100.0 [92.6 to 100.0] | 98.9 [94.3 to 100.0] | 0.0 [0.0 to 14.2] | 3.3 [0.1 to 7.2] | 1.9 [0.0 to 9.9]
  T3: PMB2001 (A56)-1:32: number analyzed (Participants) | 9 | 10 | 19 | 47 | 48 | 95 | 24 | 30 | 54
  T3: PMB2001 (A56)-1:32 | 100.0 [66.4 to 100.0] | 90.0 [55.5 to 99.7] | 94.7 [74.0 to 99.9] | 97.9 [88.7 to 99.9] | 93.8 [82.8 to 98.7] | 95.8 [89.6 to 98.8] | 0.0 [0.0 to 14.2] | 3.3 [0.1 to 17.2] | 1.9 [0.0 to 9.9]
  T3: PMB2001 (A56)-1:64: number analyzed (Participants) | 9 | 10 | 19 | 47 | 48 | 95 | 24 | 30 | 54
  T3: PMB2001 (A56)-1:64 | 100.0 [66.4 to 100.0] | 80.0 [44.4 to 97.5] | 89.5 [66.9 to 98.7] | 93.6 [82.5 to 98.7] | 85.4 [72.2 to 93.9] | 89.5 [81.5 to 94.8] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 6.6]
  T3: PMB2001 (A56)-1:128: number analyzed (Participants) | 9 | 10 | 19 | 47 | 48 | 95 | 24 | 30 | 54
  T3: PMB2001 (A56)-1:128 | 55.6 [21.2 to 86.3] | 80.0 [44.4 to 97.5] | 68.4 [43.4 to 87.4] | 89.4 [76.9 to 96.5] | 77.1 [62.7 to 88.0] | 83.2 [74.1 to 90.1] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 6.6]
  T3:PMB2948 (B24)-1:4: number analyzed (Participants) | 9 | 11 | 20 | 45 | 50 | 95 | 31 | 29 | 60
  T3:PMB2948 (B24)-1:4 | 88.9 [51.8 to 99.7] | 81.8 [48.2 to 97.7] | 85.0 [62.1 to 96.8] | 71.1 [55.7 to 83.6] | 72.0 [57.5 to 83.8] | 71.6 [61.4 to 80.4] | 3.2 [0.1 to 16.7] | 6.9 [0.8 to 22.8] | 5.0 [1.0 to 13.9]
  T3:PMB2948 (B24)-1:16: number analyzed (Participants) | 9 | 11 | 20 | 45 | 50 | 95 | 31 | 29 | 60
  T3:PMB2948 (B24)-1:16 | 88.9 [51.8 to 99.7] | 63.6 [30.8 to 89.1] | 75.0 [50.9 to 91.3] | 66.7 [51.0 to 80.0] | 68.0 [53.3 to 80.5] | 67.4 [57.0 to 76.6] | 3.2 [0.1 to 16.7] | 6.9 [0.8 to 22.8] | 5.0 [1.0 to 13.9]
  T3:PMB2948 (B24)-1:32: number analyzed (Participants) | 9 | 11 | 20 | 45 | 50 | 95 | 31 | 29 | 60
  T3:PMB2948 (B24)-1:32 | 44.4 [13.7 to 78.8] | 36.4 [10.9 to 69.2] | 40.0 [19.1 to 63.9] | 37.8 [23.8 to 53.5] | 34.0 [21.2 to 48.8] | 35.8 [26.2 to 46.3] | 3.2 [0.1 to 16.7] | 0.0 [0.0 to 11.9] | 1.7 [0.0 to 8.9]
  T3:PMB2948 (B24)-1:64: number analyzed (Participants) | 9 | 11 | 20 | 45 | 50 | 95 | 31 | 29 | 60
  T3:PMB2948 (B24)-1:64 | 11.1 [0.3 to 48.2] | 18.2 [2.3 to 51.8] | 15.0 [3.2 to 37.9] | 17.8 [8.0 to 32.1] | 10.0 [3.3 to 21.8] | 13.7 [7.5 to 22.3] | 0.0 [0.0 to 11.2] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 6.0]
  T3:PMB2948 (B24)-1:128: number analyzed (Participants) | 9 | 11 | 20 | 45 | 50 | 95 | 31 | 29 | 60
  T3:PMB2948 (B24)-1:128 | 0.0 [0.0 to 33.6] | 9.1 [0.2 to 41.3] | 5.0 [0.1 to 24.9] | 2.2 [0.1 to 11.8] | 2.0 [0.1 to 10.6] | 2.1 [0.3 to 7.4] | 0.0 [0.0 to 11.2] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 6.0]
  T3:PMB2707 (B44)-1:4: number analyzed (Participants) | 9 | 10 | 19 | 47 | 47 | 94 | 24 | 30 | 54
  T3:PMB2707 (B44)-1:4 | 88.9 [51.8 to 99.7] | 90.0 [55.5 to 99.7] | 89.5 [66.9 to 98.7] | 87.2 [74.3 to 95.2] | 87.2 [74.3 to 95.2] | 87.2 [78.8 to 93.2] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 6.6]
  T3:PMB2707 (B44)-1:16: number analyzed (Participants) | 9 | 10 | 19 | 47 | 47 | 94 | 24 | 30 | 54
  T3:PMB2707 (B44)-1:16 | 77.8 [40.0 to 97.2] | 90.0 [55.5 to 99.7] | 84.2 [60.4 to 96.6] | 87.2 [74.3 to 95.2] | 85.1 [71.7 to 93.8] | 86.2 [77.5 to 92.4] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 6.6]
  T3:PMB2707 (B44)-1:32: number analyzed (Participants) | 9 | 10 | 19 | 47 | 47 | 94 | 24 | 30 | 54
  T3:PMB2707 (B44)-1:32 | 55.6 [21.2 to 86.3] | 70.0 [34.8 to 93.3] | 63.2 [38.4 to 83.7] | 74.5 [59.7 to 86.1] | 78.7 [64.3 to 89.3] | 76.6 [66.7 to 84.7] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 6.6]
  T3:PMB2707 (B44)-1:64: number analyzed (Participants) | 9 | 10 | 19 | 47 | 47 | 94 | 24 | 30 | 54
  T3:PMB2707 (B44)-1:64 | 44.4 [13.7 to 78.8] | 30.0 [6.7 to 65.2] | 36.8 [16.3 to 61.6] | 57.4 [42.2 to 71.7] | 59.6 [44.3 to 73.6] | 58.5 [47.9 to 68.6] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 6.6]
  T3:PMB2707 (B44)-1:128: number analyzed (Participants) | 9 | 10 | 19 | 47 | 47 | 94 | 24 | 30 | 54
  T3:PMB2707 (B44)-1:128 | 22.2 [2.8 to 60.0] | 20.0 [2.5 to 55.6] | 21.1 [6.1 to 45.6] | 29.8 [17.3 to 44.9] | 34.0 [20.9 to 49.3] | 31.9 [22.7 to 42.3] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 6.6]
  T4: PMB80 (A22): 1: 4: number analyzed (Participants) | 10 | 10 | 20 | 46 | 51 | 97 | 30 | 28 | 58
  T4: PMB80 (A22): 1: 4 | 20.0 [2.5 to 55.6] | 0.0 [0.0 to 30.8] | 10.0 [1.2 to 31.7] | 17.4 [7.8 to 31.4] | 7.8 [2.2 to 18.9] | 12.4 [6.6 to 20.6] | 0.0 [0.0 to 11.6] | 7.1 [0.9 to 23.5] | 3.4 [0.4 to 11.9]
  T4: PMB80 (A22): 1: 8: number analyzed (Participants) | 10 | 10 | 20 | 46 | 51 | 97 | 30 | 28 | 58
  T4: PMB80 (A22): 1: 8 | 20.0 [2.5 to 55.6] | 0.0 [0.0 to 30.8] | 10.0 [1.2 to 31.7] | 17.4 [7.8 to 31.4] | 7.8 [2.2 to 18.9] | 12.4 [6.6 to 20.6] | 0.0 [0.0 to 11.6] | 7.1 [0.9 to 23.5] | 3.4 [0.4 to 11.9]
  T4: PMB80 (A22): 1: 16: number analyzed (Participants) | 10 | 10 | 20 | 46 | 51 | 97 | 30 | 28 | 58
  T4: PMB80 (A22): 1: 16 | 20.0 [2.5 to 55.6] | 0.0 [0.0 to 30.8] | 10.0 [1.2 to 31.7] | 17.4 [7.8 to 31.4] | 7.8 [2.2 to 18.9] | 12.4 [6.6 to 20.6] | 0.0 [0.0 to 11.6] | 7.1 [0.9 to 23.5] | 3.4 [0.4 to 11.9]
  T4: PMB80 (A22): 1: 32: number analyzed (Participants) | 10 | 10 | 20 | 46 | 51 | 97 | 30 | 28 | 58
  T4: PMB80 (A22): 1: 32 | 10.0 [0.3 to 44.5] | 0.0 [0.0 to 30.8] | 5.0 [0.1 to 24.9] | 15.2 [6.3 to 28.9] | 5.9 [1.2 to 16.2] | 10.3 [5.1 to 18.1] | 0.0 [0.0 to 11.6] | 3.6 [0.1 to 18.3] | 1.7 [0.0 to 9.2]
  T4: PMB80 (A22): 1: 64: number analyzed (Participants) | 10 | 10 | 20 | 46 | 51 | 97 | 30 | 28 | 58
  T4: PMB80 (A22): 1: 64 | 10.0 [0.3 to 44.5] | 0.0 [0.0 to 30.8] | 5.0 [0.1 to 24.9] | 6.5 [1.4 to 17.9] | 2.0 [0.0 to 10.4] | 4.1 [1.1 to 10.2] | 0.0 [0.0 to 11.6] | 3.6 [0.1 to 18.3] | 1.7 [0.0 to 9.2]
  T4: PMB80 (A22): 1: 128: number analyzed (Participants) | 10 | 10 | 20 | 46 | 51 | 97 | 30 | 28 | 58
  T4: PMB80 (A22): 1: 128 | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 16.8] | 2.2 [0.1 to 11.5] | 2.0 [0.0 to 10.4] | 2.1 [0.3 to 7.3] | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 12.3] | 0.0 [0.0 to 6.2]
  T4: PMB2001 (A56): 1:4: number analyzed (Participants) | 8 | 10 | 18 | 41 | 47 | 88 | 24 | 28 | 52
  T4: PMB2001 (A56): 1:4 | 62.5 [24.5 to 91.5] | 80.0 [44.4 to 97.5] | 72.2 [46.5 to 90.3] | 65.9 [49.4 to 79.9] | 63.8 [48.5 to 77.3] | 64.8 [53.9 to 74.7] | 4.2 [0.1 to 21.1] | 3.6 [0.1 to 18.3] | 3.8 [0.5 to 13.2]
  T4: PMB2001 (A56): 1:8: number analyzed (Participants) | 8 | 10 | 18 | 41 | 47 | 88 | 24 | 28 | 52
  T4: PMB2001 (A56): 1:8 | 37.5 [8.5 to 75.5] | 80.0 [44.4 to 97.5] | 61.1 [35.7 to 82.7] | 61.0 [44.5 to 75.8] | 57.4 [42.2 to 71.7] | 59.1 [48.1 to 69.5] | 4.2 [0.1 to 21.1] | 3.6 [0.1 to 18.3] | 3.8 [0.5 to 13.2]
  T4: PMB2001 (A56): 1:16: number analyzed (Participants) | 8 | 10 | 18 | 41 | 47 | 88 | 24 | 28 | 52
  T4: PMB2001 (A56): 1:16 | 25.0 [3.2 to 65.1] | 80.0 [44.4 to 97.5] | 55.6 [30.8 to 78.5] | 58.5 [42.1 to 73.7] | 44.7 [30.2 to 59.9] | 51.1 [40.2 to 61.9] | 0.0 [0.0 to 14.2] | 3.6 [0.1 to 18.3] | 1.9 [0.0 to 10.3]
  T4: PMB2001 (A56): 1:32: number analyzed (Participants) | 8 | 10 | 18 | 41 | 47 | 88 | 24 | 28 | 52
  T4: PMB2001 (A56): 1:32 | 25.0 [3.2 to 65.1] | 60.0 [26.2 to 87.8] | 44.5 [21.5 to 69.2] | 34.1 [20.1 to 50.6] | 31.9 [19.1 to 47.1] | 33.0 [23.3 to 43.8] | 0.0 [0.0 to 14.2] | 3.6 [0.1 to 18.3] | 1.9 [0.0 to 10.3]
  T4: PMB2001 (A56): 1:64: number analyzed (Participants) | 8 | 10 | 18 | 41 | 47 | 88 | 24 | 28 | 52
  T4: PMB2001 (A56): 1:64 | 0.0 [0.0 to 36.9] | 40.0 [12.2 to 73.8] | 22.2 [6.4 to 47.6] | 14.6 [5.6 to 29.2] | 21.3 [10.7 to 35.7] | 18.2 [10.8 to 27.8] | 0.0 [0.0 to 14.2] | 3.6 [0.1 to 18.3] | 1.9 [0.0 to 10.3]
  T4: PMB2001 (A56): 1:128: number analyzed (Participants) | 8 | 10 | 18 | 41 | 47 | 88 | 24 | 28 | 52
  T4: PMB2001 (A56): 1:128 | 0.0 [0.0 to 36.9] | 20.0 [2.5 to 55.6] | 11.1 [1.4 to 34.7] | 4.9 [0.6 to 16.5] | 8.5 [2.4 to 20.4] | 6.8 [2.5 to 14.3] | 0.0 [0.0 to 14.2] | 3.6 [0.1 to 18.3] | 1.9 [0.0 to 10.3]
  T4: PMB2948 (B24): 1: 4: number analyzed (Participants) | 10 | 10 | 20 | 46 | 51 | 97 | 30 | 28 | 58
  T4: PMB2948 (B24): 1: 4 | 20.0 [2.5 to 55.6] | 10.0 [0.3 to 44.5] | 15.0 [3.2 to 37.9] | 10.9 [3.6 to 23.6] | 15.7 [7.0 to 28.6] | 13.4 [7.3 to 21.8] | 3.3 [0.1 to 17.2] | 3.6 [0.1 to 18.3] | 3.4 [0.4 to 11.9]
  T4: PMB2948 (B24): 1: 8: number analyzed (Participants) | 10 | 10 | 20 | 46 | 51 | 97 | 30 | 28 | 58
  T4: PMB2948 (B24): 1: 8 | 20.0 [2.5 to 55.6] | 10.0 [0.3 to 44.5] | 15.0 [3.2 to 37.9] | 8.7 [2.4 to 20.8] | 11.8 [4.4 to 23.9] | 10.3 [5.1 to 18.1] | 3.3 [0.1 to 17.2] | 3.6 [0.1 to 18.3] | 3.4 [0.4 to 11.9]
  T4: PMB2948 (B24): 1: 16: number analyzed (Participants) | 10 | 10 | 20 | 46 | 51 | 97 | 30 | 28 | 58
  T4: PMB2948 (B24): 1: 16 | 10.0 [0.3 to 44.5] | 10.0 [0.3 to 44.5] | 10.0 [1.2 to 31.7] | 6.5 [1.4 to 17.9] | 11.8 [4.4 to 23.9] | 9.3 [4.3 to 16.9] | 0.0 [0.0 to 11.6] | 3.6 [0.1 to 18.3] | 1.7 [0.0 to 9.2]
  T4: PMB2948 (B24): 1: 32: number analyzed (Participants) | 10 | 10 | 20 | 46 | 51 | 97 | 30 | 28 | 58
  T4: PMB2948 (B24): 1: 32 | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 16.8] | 0.0 [0.0 to 7.7] | 3.9 [0.5 to 13.5] | 2.1 [0.3 to 7.3] | 0.0 [0.0 to 11.6] | 3.6 [0.1 to 18.3] | 1.7 [0.0 to 9.2]
  T4: PMB2948 (B24): 1: 64: number analyzed (Participants) | 10 | 10 | 20 | 46 | 51 | 97 | 30 | 28 | 58
  T4: PMB2948 (B24): 1: 64 | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 16.8] | 0.0 [0.0 to 7.7] | 2.0 [0.0 to 10.4] | 1.0 [0.0 to 5.6] | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 12.3] | 0.0 [0.0 to 6.2]
  T4: PMB2948 (B24): 1: 128: number analyzed (Participants) | 10 | 10 | 20 | 46 | 51 | 97 | 30 | 28 | 58
  T4: PMB2948 (B24): 1: 128 | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 16.8] | 0.0 [0.0 to 7.7] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 3.7] | 0.0 [0.0 to 11.6] | 0.0 [0.0 to 12.3] | 0.0 [0.0 to 6.2]
  T4: PMB2707 (B44): 1: 4: number analyzed (Participants) | 8 | 8 | 16 | 43 | 46 | 89 | 24 | 29 | 53
  T4: PMB2707 (B44): 1: 4 | 12.5 [0.3 to 52.7] | 37.5 [8.5 to 75.5] | 25.0 [7.3 to 52.4] | 44.2 [29.1 to 60.1] | 47.8 [32.9 to 63.1] | 46.1 [35.4 to 57.0] | 4.2 [0.1 to 21.1] | 0.0 [0.0 to 11.9] | 1.9 [0.0 to 10.1]
  T4: PMB2707 (B44): 1: 8: number analyzed (Participants) | 8 | 8 | 16 | 43 | 46 | 89 | 24 | 29 | 53
  T4: PMB2707 (B44): 1: 8 | 12.5 [0.3 to 52.7] | 37.5 [8.5 to 75.5] | 25.0 [7.3 to 52.4] | 39.5 [25.0 to 55.6] | 41.3 [27.0 to 56.8] | 40.4 [30.2 to 51.4] | 4.2 [0.1 to 21.1] | 0.0 [0.0 to 11.9] | 1.9 [0.0 to 10.1]
  T4: PMB2707 (B44): 1: 16: number analyzed (Participants) | 8 | 8 | 16 | 43 | 46 | 89 | 24 | 29 | 53
  T4: PMB2707 (B44): 1: 16 | 12.5 [0.3 to 52.7] | 25.0 [3.2 to 65.1] | 18.8 [4.0 to 45.6] | 34.9 [21.0 to 50.9] | 32.6 [19.5 to 48.0] | 33.7 [24.0 to 44.5] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 6.7]
  T4: PMB2707 (B44): 1: 32: number analyzed (Participants) | 8 | 8 | 16 | 43 | 46 | 89 | 24 | 29 | 53
  T4: PMB2707 (B44): 1: 32 | 0.0 [0.0 to 36.9] | 12.5 [0.3 to 52.7] | 6.3 [0.2 to 30.2] | 11.6 [3.9 to 25.1] | 10.9 [3.6 to 23.6] | 11.2 [5.5 to 19.7] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 6.7]
  T4: PMB2707 (B44): 1: 64: number analyzed (Participants) | 8 | 8 | 16 | 43 | 46 | 89 | 24 | 29 | 53
  T4: PMB2707 (B44): 1: 64 | 0.0 [0.0 to 36.9] | 12.5 [0.3 to 52.7] | 6.3 [0.2 to 30.2] | 9.3 [2.6 to 22.1] | 2.2 [0.1 to 11.5] | 5.6 [1.8 to 12.6] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 6.7]
  T4: PMB2707 (B44): 1: 128: number analyzed (Participants) | 8 | 8 | 16 | 43 | 46 | 89 | 24 | 29 | 53
  T4: PMB2707 (B44): 1: 128 | 0.0 [0.0 to 36.9] | 12.5 [0.3 to 52.7] | 6.3 [0.2 to 30.2] | 2.3 [0.1 to 12.3] | 0.0 [0.0 to 7.7] | 1.1 [0.0 to 6.1] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 6.7]
  T5: PMB80 (A22): 1:4: number analyzed (Participants) | 10 | 11 | 21 | 45 | 50 | 95 | 27 | 28 | 55
  T5: PMB80 (A22): 1:4 | 10.0 [0.3 to 44.5] | 18.2 [2.3 to 51.8] | 14.3 [3.0 to 36.3] | 13.3 [5.1 to 26.8] | 6.0 [1.3 to 16.5] | 9.5 [4.4 to 17.2] | 3.7 [0.1 to 19.0] | 3.6 [0.1 to 18.3] | 3.6 [0.4 to 12.5]
  T5: PMB80 (A22): 1: 8: number analyzed (Participants) | 10 | 11 | 21 | 45 | 50 | 95 | 27 | 28 | 55
  T5: PMB80 (A22): 1: 8 | 10.0 [0.3 to 44.5] | 18.2 [2.3 to 51.8] | 14.3 [3.0 to 36.3] | 11.1 [3.7 to 24.1] | 4.0 [0.5 to 13.7] | 7.4 [3.0 to 14.6] | 3.7 [0.1 to 19.0] | 0.0 [0.0 to 12.3] | 1.8 [0.0 to 9.7]
  T5: PMB80 (A22): 1: 16: number analyzed (Participants) | 10 | 11 | 21 | 45 | 50 | 95 | 27 | 28 | 55
  T5: PMB80 (A22): 1: 16 | 10.0 [0.3 to 44.5] | 18.2 [2.3 to 51.8] | 14.3 [3.0 to 36.3] | 8.9 [2.5 to 21.2] | 4.0 [0.5 to 13.7] | 6.3 [2.4 to 13.22] | 3.7 [0.1 to 19.0] | 0.0 [0.0 to 12.3] | 1.8 [0.0 to 9.7]
  T5: PMB80 (A22): 1: 32: number analyzed (Participants) | 10 | 11 | 21 | 45 | 50 | 95 | 27 | 28 | 55
  T5: PMB80 (A22): 1: 32 | 0.0 [0.0 to 30.8] | 9.1 [0.2 to 41.3] | 4.8 [0.1 to 23.8] | 4.4 [0.5 to 15.1] | 4.0 [0.5 to 13.7] | 4.2 [1.2 to 10.4] | 0.0 [0.0 to 12.8] | 0.0 [0.0 to 12.3] | 0.0 [0.0 to 6.5]
  T5: PMB80 (A22): 1: 64: number analyzed (Participants) | 10 | 11 | 21 | 45 | 50 | 95 | 27 | 28 | 55
  T5: PMB80 (A22): 1: 64 | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 16.1] | 2.2 [0.1 to 11.8] | 2.0 [0.1 to 10.6] | 2.1 [0.3 to 7.4] | 0.0 [0.0 to 12.8] | 0.0 [0.0 to 12.3] | 0.0 [0.0 to 6.5]
  T5: PMB80 (A22): 1: 128: number analyzed (Participants) | 10 | 11 | 21 | 45 | 50 | 95 | 27 | 28 | 55
  T5: PMB80 (A22): 1: 128 | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 7.9] | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 3.8] | 0.0 [0.0 to 12.8] | 0.0 [0.0 to 12.3] | 0.0 [0.0 to 6.5]
  T5: PMB2001 (A56): 1: 4: number analyzed (Participants) | 9 | 7 | 16 | 45 | 48 | 93 | 23 | 30 | 53
  T5: PMB2001 (A56): 1: 4 | 33.3 [7.5 to 70.1] | 85.7 [42.1 to 99.6] | 56.3 [29.9 to 80.2] | 53.3 [37.9 to 68.3] | 52.1 [37.2 to 66.7] | 52.7 [42.1 to 63.1] | 8.7 [1.1 to 28.0] | 10.0 [2.1 to 26.5] | 9.4 [3.1 to 20.7]
  T5: PMB2001 (A56): 1: 8: number analyzed (Participants) | 9 | 7 | 16 | 45 | 48 | 93 | 23 | 30 | 53
  T5: PMB2001 (A56): 1: 8 | 33.3 [7.5 to 70.1] | 85.7 [42.1 to 99.6] | 56.3 [29.9 to 80.2] | 40.0 [25.7 to 55.7] | 37.5 [24.0 to 52.6] | 38.7 [28.8 to 49.4] | 0.0 [0.0 to 14.8] | 10.0 [2.1 to 26.5] | 5.7 [1.2 to 15.7]
  T5: PMB2001 (A56): 1: 16: number analyzed (Participants) | 9 | 7 | 16 | 45 | 48 | 93 | 23 | 30 | 53
  T5: PMB2001 (A56): 1: 16 | 33.3 [7.5 to 70.1] | 85.7 [42.1 to 99.6] | 56.3 [29.9 to 80.2] | 26.7 [14.6 to 41.9] | 31.3 [18.7 to 46.3] | 29.0 [20.1 to 39.4] | 0.0 [0.0 to 14.8] | 10.0 [2.1 to 26.5] | 5.7 [1.2 to 15.7]
  T5: PMB2001 (A56): 1: 32: number analyzed (Participants) | 9 | 7 | 16 | 45 | 48 | 93 | 23 | 30 | 53
  T5: PMB2001 (A56): 1: 32 | 22.2 [2.8 to 60.0] | 71.4 [29.0 to 96.3] | 43.8 [19.8 to 70.1] | 17.8 [8.0 to 32.1] | 20.8 [10.5 to 35.0] | 19.4 [11.9 to 28.9] | 0.0 [0.0 to 14.8] | 10.0 [2.1 to 26.5] | 5.7 [1.2 to 15.7]
  T5: PMB2001 (A56): 1: 64: number analyzed (Participants) | 9 | 7 | 16 | 45 | 48 | 93 | 23 | 30 | 53
  T5: PMB2001 (A56): 1: 64 | 22.2 [2.8 to 60.0] | 42.9 [9.9 to 81.6] | 31.3 [11.0 to 58.7] | 8.9 [2.5 to 21.2] | 12.5 [4.7 to 25.2] | 10.8 [5.3 to 18.9] | 0.0 [0.0 to 14.8] | 6.7 [0.8 to 22.1] | 3.8 [0.5 to 13.0]
  T5: PMB2001 (A56): 1: 128: number analyzed (Participants) | 9 | 7 | 16 | 45 | 48 | 93 | 23 | 30 | 53
  T5: PMB2001 (A56): 1: 128 | 0.0 [0.0 to 33.6] | 28.6 [3.7 to 71.0] | 12.5 [1.6 to 38.3] | 4.4 [0.5 to 15.1] | 0.0 [0.0 to 7.4] | 2.2 [0.3 to 7.6] | 0.0 [0.0 to 14.8] | 3.3 [0.1 to 17.2] | 1.9 [0.0 to 10.1]
  T5: PMB2948 (B24): 1: 4: number analyzed (Participants) | 10 | 11 | 21 | 44 | 49 | 93 | 27 | 28 | 55
  T5: PMB2948 (B24): 1: 4 | 0.0 [0.0 to 30.8] | 27.3 [6.0 to 61.0] | 14.3 [3.0 to 36.3] | 2.3 [0.1 to 12.0] | 6.1 [1.3 to 16.9] | 4.3 [1.2 to 10.6] | 0.0 [0.0 to 12.8] | 7.1 [0.9 to 23.5] | 3.6 [0.4 to 12.5]
  T5: PMB2948 (B24): 1: 8: number analyzed (Participants) | 10 | 11 | 21 | 44 | 49 | 93 | 27 | 28 | 55
  T5: PMB2948 (B24): 1: 8 | 0.0 [0.0 to 30.8] | 18.2 [2.3 to 51.8] | 9.5 [1.2 to 30.4] | 2.3 [0.1 to 12.0] | 4.1 [0.5 to 14.0] | 3.2 [0.7 to 9.1] | 0.0 [0.0 to 12.8] | 7.1 [0.9 to 23.5] | 3.6 [0.4 to 12.5]
  T5: PMB2948 (B24): 1: 16: number analyzed (Participants) | 10 | 11 | 21 | 44 | 49 | 93 | 27 | 28 | 55
  T5: PMB2948 (B24): 1: 16 | 0.0 [0.0 to 30.8] | 18.2 [2.3 to 51.8] | 9.5 [1.2 to 30.4] | 0.0 [0.0 to 8.0] | 2.0 [0.1 to 10.9] | 1.1 [0.0 to 5.8] | 0.0 [0.0 to 12.8] | 7.1 [0.9 to 23.5] | 3.6 [0.4 to 12.5]
  T5: PMB2948 (B24): 1: 32: number analyzed (Participants) | 10 | 11 | 21 | 44 | 49 | 93 | 27 | 28 | 55
  T5: PMB2948 (B24): 1: 32 | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 8.0] | 2.0 [0.1 to 10.9] | 1.1 [0.0 to 5.8] | 0.0 [0.0 to 12.8] | 3.6 [0.1 to 18.3] | 1.8 [0.0 to 9.7]
  T5: PMB2948 (B24): 1: 64: number analyzed (Participants) | 10 | 11 | 21 | 44 | 49 | 93 | 27 | 28 | 55
  T5: PMB2948 (B24): 1: 64 | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 8.0] | 2.0 [0.1 to 10.9] | 1.1 [0.0 to 5.8] | 0.0 [0.0 to 12.8] | 3.6 [0.1 to 18.3] | 1.8 [0.0 to 9.7]
  T5: PMB2948 (B24): 1: 128: number analyzed (Participants) | 10 | 11 | 21 | 44 | 49 | 93 | 27 | 28 | 55
  T5: PMB2948 (B24): 1: 128 | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 8.0] | 2.0 [0.1 to 10.9] | 1.1 [0.0 to 5.8] | 0.0 [0.0 to 12.8] | 0.0 [0.0 to 12.3] | 0.0 [0.0 to 6.5]
  T5: PMB2707 (B44): 1:4: number analyzed (Participants) | 9 | 7 | 16 | 43 | 47 | 90 | 22 | 29 | 51
  T5: PMB2707 (B44): 1:4 | 11.1 [0.3 to 48.2] | 14.3 [0.4 to 57.9] | 12.5 [1.6 to 38.3] | 20.9 [10.0 to 36.0] | 21.3 [10.7 to 35.7] | 21.1 [13.2 to 31.0] | 4.5 [0.1 to 22.8] | 3.4 [0.1 to 17.8] | 3.9 [0.5 to 13.5]
  T5: PMB2707 (B44): 1:8: number analyzed (Participants) | 9 | 7 | 16 | 43 | 47 | 90 | 22 | 29 | 51
  T5: PMB2707 (B44): 1:8 | 11.1 [0.3 to 48.2] | 14.3 [0.4 to 57.9] | 12.5 [1.6 to 38.3] | 18.6 [8.4 to 33.4] | 17.0 [7.6 to 30.8] | 17.8 [10.5 to 27.3] | 0.0 [0.0 to 15.4] | 3.4 [0.1 to 17.8] | 2.0 [0.0 to 10.4]
  T5: PMB2707 (B44): 1:16: number analyzed (Participants) | 9 | 7 | 16 | 43 | 47 | 90 | 22 | 29 | 51
  T5: PMB2707 (B44): 1:16 | 0.0 [0.0 to 33.6] | 14.3 [0.4 to 57.9] | 6.3 [0.2 to 30.2] | 16.3 [6.8 to 30.7] | 8.5 [2.4 to 20.4] | 12.2 [6.3 to 20.8] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 7.0]
  T5: PMB2707 (B44): 1:32: number analyzed (Participants) | 9 | 7 | 16 | 43 | 47 | 90 | 22 | 29 | 51
  T5: PMB2707 (B44): 1:32 | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 20.6] | 4.7 [0.6 to 15.8] | 4.3 [0.5 to 14.5] | 4.4 [1.2 to 11.0] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 7.0]
  T5: PMB2707 (B44): 1:64: number analyzed (Participants) | 9 | 7 | 16 | 43 | 47 | 90 | 22 | 29 | 51
  T5: PMB2707 (B44): 1:64 | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 20.6] | 2.3 [0.1 to 12.3] | 2.1 [0.1 to 11.3] | 2.2 [0.3 to 7.8] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 7.0]
  T5: PMB2707 (B44): 1:128: number analyzed (Participants) | 9 | 7 | 16 | 43 | 47 | 90 | 22 | 29 | 51
  T5: PMB2707 (B44): 1:128 | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 8.2] | 0.0 [0.0 to 7.5] | 0.0 [0.0 to 4.0] | 0.0 [0.0 to 15.4] | 0.0 [0.0 to 11.9] | 0.0 [0.0 to 7.0]
  T6: PMB80 (A22): 1:4: number analyzed (Participants) | 10 | 9 | 19 | 34 | 47 | 81 | 0 | 0 | 0
  T6: PMB80 (A22): 1:4 | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 17.6] | 8.8 [1.9 to 23.7] | 2.1 [0.1 to 11.3] | 4.9 [1.4 to 12.2] |  |  |
  T6: PMB80 (A22): 1:8: number analyzed (Participants) | 10 | 9 | 19 | 34 | 47 | 81 | 0 | 0 | 0
  T6: PMB80 (A22): 1:8 | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 17.6] | 5.9 [0.7 to 19.7] | 2.1 [0.1 to 11.3] | 3.7 [0.8 to 10.4] |  |  |
  T6: PMB80 (A22): 1:16: number analyzed (Participants) | 10 | 9 | 19 | 34 | 47 | 81 | 0 | 0 | 0
  T6: PMB80 (A22): 1:16 | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 17.6] | 5.9 [0.7 to 19.7] | 2.1 [0.1 to 11.3] | 3.7 [0.8 to 10.4] |  |  |
  T6: PMB80 (A22): 1:32: number analyzed (Participants) | 10 | 9 | 19 | 34 | 47 | 81 | 0 | 0 | 0
  T6: PMB80 (A22): 1:32 | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 17.6] | 5.9 [0.7 to 19.7] | 2.1 [0.1 to 11.3] | 3.7 [0.8 to 10.4] |  |  |
  T6: PMB80 (A22): 1:64: number analyzed (Participants) | 10 | 9 | 19 | 34 | 47 | 81 | 0 | 0 | 0
  T6: PMB80 (A22): 1:64 | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 17.6] | 2.9 [0.1 to 15.3] | 2.1 [0.1 to 11.3] | 2.5 [0.3 to 8.6] |  |  |
  T6: PMB80 (A22): 1:128: number analyzed (Participants) | 10 | 9 | 19 | 34 | 47 | 81 | 0 | 0 | 0
  T6: PMB80 (A22): 1:128 | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 17.6] | 0.0 [0.0 to 10.3] | 0.0 [0.0 to 7.5] | 0.0 [0.0 to 4.5] |  |  |
  T6: PMB2001 (A56): 1:4: number analyzed (Participants) | 9 | 8 | 17 | 39 | 40 | 79 | 0 | 0 | 0
  T6: PMB2001 (A56): 1:4 | 22.2 [2.8 to 60.0] | 75.0 [34.9 to 96.8] | 47.1 [23.0 to 72.2] | 20.5 [9.3 to 36.5] | 30.0 [16.6 to 46.5] | 25.3 [16.2 to 36.4] |  |  |
  T6: PMB2001 (A56): 1:8: number analyzed (Participants) | 9 | 8 | 17 | 39 | 40 | 79 | 0 | 0 | 0
  T6: PMB2001 (A56): 1:8 | 11.1 [0.3 to 48.2] | 75.0 [34.9 to 96.8] | 41.2 [18.4 to 67.1] | 15.4 [5.9 to 30.5] | 30.0 [16.6 to 46.5] | 22.8 [14.1 to 33.6] |  |  |
  T6: PMB2001 (A56): 1:16: number analyzed (Participants) | 9 | 8 | 17 | 39 | 40 | 79 | 0 | 0 | 0
  T6: PMB2001 (A56): 1:16 | 11.1 [0.3 to 48.2] | 75.0 [34.9 to 96.8] | 41.2 [18.4 to 67.1] | 10.3 [2.9 to 24.2] | 27.5 [14.6 to 43.9] | 19.0 [11.0 to 29.4] |  |  |
  T6: PMB2001 (A56): 1:32: number analyzed (Participants) | 9 | 8 | 17 | 39 | 40 | 79 | 0 | 0 | 0
  T6: PMB2001 (A56): 1:32 | 11.1 [0.3 to 48.2] | 50.0 [15.7 to 84.3] | 29.4 [10.3 to 56.0] | 2.6 [0.1 to 13.5] | 12.5 [4.2 to 26.8] | 7.6 [2.8 to 15.8] |  |  |
  T6: PMB2001 (A56): 1:64: number analyzed (Participants) | 9 | 8 | 17 | 39 | 40 | 79 | 0 | 0 | 0
  T6: PMB2001 (A56): 1:64 | 11.1 [0.3 to 48.2] | 0.0 [0.0 to 36.9] | 5.9 [0.1 to 28.7] | 2.6 [0.1 to 13.5] | 7.5 [1.6 to 20.4] | 5.1 [1.4 to 12.5] |  |  |
  T6: PMB2001 (A56): 1:128: number analyzed (Participants) | 9 | 8 | 17 | 39 | 40 | 79 | 0 | 0 | 0
  T6: PMB2001 (A56): 1:128 | 11.1 [0.3 to 48.2] | 0.0 [0.0 to 36.9] | 5.9 [0.1 to 28.7] | 2.6 [0.1 to 13.5] | 5.0 [0.6 to 16.9] | 3.8 [0.8 to 10.7] |  |  |
  T6: PMB2948 (B24): 1: 4: number analyzed (Participants) | 10 | 9 | 19 | 34 | 48 | 82 | 0 | 0 | 0
  T6: PMB2948 (B24): 1: 4 | 0.0 [0.0 to 30.8] | 11.1 [0.3 to 48.2] | 5.3 [0.1 to 26.0] | 8.8 [1.9 to 23.7] | 0.0 [0.0 to 7.4] | 3.7 [0.8 to 10.3] |  |  |
  T6: PMB2948 (B24): 1: 8: number analyzed (Participants) | 10 | 9 | 19 | 34 | 48 | 82 | 0 | 0 | 0
  T6: PMB2948 (B24): 1: 8 | 0.0 [0.0 to 30.8] | 11.1 [0.3 to 48.2] | 5.3 [0.1 to 26.0] | 8.8 [1.9 to 23.7] | 0.0 [0.0 to 7.4] | 3.7 [0.8 to 10.3] |  |  |
  T6: PMB2948 (B24): 1: 16: number analyzed (Participants) | 10 | 9 | 19 | 34 | 48 | 82 | 0 | 0 | 0
  T6: PMB2948 (B24): 1: 16 | 0.0 [0.0 to 30.8] | 11.1 [0.3 to 48.2] | 5.3 [0.1 to 26.0] | 5.9 [0.7 to 19.7] | 0.0 [0.0 to 7.4] | 2.4 [0.3 to 8.5] |  |  |
  T6: PMB2948 (B24): 1: 32: number analyzed (Participants) | 10 | 9 | 19 | 34 | 48 | 82 | 0 | 0 | 0
  T6: PMB2948 (B24): 1: 32 | 0.0 [0.0 to 30.8] | 11.1 [0.3 to 48.2] | 5.3 [0.1 to 26.0] | 5.9 [0.7 to 19.7] | 0.0 [0.0 to 7.4] | 2.4 [0.3 to 8.5] |  |  |
  T6: PMB2948 (B24): 1: 64: number analyzed (Participants) | 10 | 9 | 19 | 34 | 48 | 82 | 0 | 0 | 0
  T6: PMB2948 (B24): 1: 64 | 0.0 [0.0 to 30.8] | 11.1 [0.3 to 48.2] | 5.3 [0.1 to 26.0] | 5.9 [0.7 to 19.7] | 0.0 [0.0 to 7.4] | 2.4 [0.3 to 8.5] |  |  |
  T6: PMB2948 (B24): 1: 128: number analyzed (Participants) | 10 | 9 | 19 | 34 | 48 | 82 | 0 | 0 | 0
  T6: PMB2948 (B24): 1: 128 | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 17.6] | 2.9 [0.1 to 15.3] | 0.0 [0.0 to 7.4] | 1.2 [0.0 to 6.6] |  |  |
  T6: PMB2707 (B44): 1: 4: number analyzed (Participants) | 9 | 8 | 17 | 39 | 41 | 80 | 0 | 0 | 0
  T6: PMB2707 (B44): 1: 4 | 0.0 [0.0 to 33.6] | 25.0 [3.2 to 65.1] | 11.8 [1.5 to 36.4] | 15.4 [5.9 to 30.5] | 12.2 [4.1 to 26.2] | 13.8 [7.1 to 23.3] |  |  |
  T6: PMB2707 (B44): 1: 8: number analyzed (Participants) | 9 | 8 | 17 | 39 | 41 | 80 | 0 | 0 | 0
  T6: PMB2707 (B44): 1: 8 | 0.0 [0.0 to 33.6] | 25.0 [3.2 to 65.1] | 11.8 [1.5 to 36.4] | 12.8 [4.3 to 27.4] | 12.2 [4.1 to 26.2] | 12.5 [6.2 to 21.8] |  |  |
  T6: PMB2707 (B44): 1: 16: number analyzed (Participants) | 9 | 8 | 17 | 39 | 41 | 80 | 0 | 0 | 0
  T6: PMB2707 (B44): 1: 16 | 0.0 [0.0 to 33.6] | 12.5 [0.3 to 52.7] | 5.9 [0.1 to 28.7] | 7.7 [1.6 to 20.9] | 9.8 [2.7 to 23.1] | 8.8 [3.6 to 17.2] |  |  |
  T6: PMB2707 (B44): 1: 32: number analyzed (Participants) | 9 | 8 | 17 | 39 | 41 | 80 | 0 | 0 | 0
  T6: PMB2707 (B44): 1: 32 | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 19.5] | 5.1 [0.6 to 17.3] | 2.4 [0.1 to 12.9] | 3.8 [0.8 to 10.6] |  |  |
  T6: PMB2707 (B44): 1: 64: number analyzed (Participants) | 9 | 8 | 17 | 39 | 41 | 80 | 0 | 0 | 0
  T6: PMB2707 (B44): 1: 64 | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 9.0] | 2.4 [0.1 to 12.9] | 1.3 [0.0 to 6.8] |  |  |
  T6: PMB2707 (B44): 1: 128: number analyzed (Participants) | 9 | 8 | 17 | 39 | 41 | 80 | 0 | 0 | 0
  T6: PMB2707 (B44): 1: 128 | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 9.0] | 2.4 [0.1 to 12.9] | 1.3 [0.0 to 6.8] |  |  |

18. Secondary Outcome: Serum Bactericidal Assay Using Human Complement (hSBA) Geometric Mean Titers (GMTs) for Each of the 4 Primary Test Strains
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: 60-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 1: 60-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 1: 60- mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 2: 120-µg Bivalent rLP2086 (>=12 Months to <18 Months) | Group 2: 120-µg Bivalent rLP2086 (>=18 Months to <24 Months) | Group 2: 120-mcg Bivalent rLP2086 (>=12 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <18 Months) | Group 3: HAV/Saline (>=18 Months to <24 Months) | Group 3: HAV/Saline (>=12 Months to <24 Months): Stage 1
Number analyzed (Participants) | 10 | 11 | 21 | 47 | 51 | 97 | 31 | 30 | 61
titer
  T1:PMB80 (A22): number analyzed (Participants) | 9 | 11 | 20 | 46 | 51 | 97 | 31 | 30 | 61
  T1:PMB80 (A22) | 8.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 8.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 8.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 8.5 [7.5 to 9.6] | 8.3 [7.8 to 8.9] | 8.4 [7.9 to 9.0] | 8.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 8.2 [7.8 to 8.6] | 8.1 [7.9 to 8.3]
  T1: PMB2001 (A56): number analyzed (Participants) | 9 | 10 | 19 | 46 | 49 | 95 | 24 | 29 | 53
  T1: PMB2001 (A56) | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.2 [3.8 to 4.5] | 4.1 [3.9 to 4.3] | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means.
  T1: PMB2948 (B24): number analyzed (Participants) | 10 | 11 | 21 | 46 | 51 | 97 | 31 | 30 | 61
  T1: PMB2948 (B24) | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.8 [3.2 to 7.4] | 4.4 [3.6 to 5.4] | 4.1 [3.9 to 4.4] | 4.1 [3.9 to 4.3] | 4.1 [4.0 to 4.3] | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.4 [3.6 to 5.3] | 4.2 [3.8 to 4.6]
  T1: PMB2707 (B44): number analyzed (Participants) | 9 | 10 | 19 | 46 | 49 | 95 | 24 | 30 | 54
  T1: PMB2707 (B44) | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.1 [3.9 to 4.2] | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.0 [4.0 to 4.1] | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means.
  T2: PMB80 (A22): number analyzed (Participants) | 10 | 9 | 19 | 45 | 50 | 95 | 30 | 29 | 59
  T2: PMB80 (A22) | 42.2 [22.6 to 79.1] | 23.5 [10.1 to 54.9] | 32.0 [19.7 to 52.0] | 24.6 [17.8 to 34.2] | 36.8 [26.9 to 50.3] | 30.4 [24.3 to 38.1] | 8.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 8.6 [7.4 to 10.0] | 8.3 [7.7 to 8.9]
  T2: PMB2001 (A56): number analyzed (Participants) | 9 | 10 | 19 | 47 | 48 | 95 | 23 | 29 | 52
  T2: PMB2001 (A56) | 101.6 [64.0 to 161.2] | 68.6 [28.2 to 166.8] | 82.6 [51.4 to 129.9] | 117.2 [89.7 to 153.0] | 104.6 [80.4 to 136.0] | 110.6 [92.0 to 133.0] | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means.
  T2: PMB2948 (B24): number analyzed (Participants) | 10 | 9 | 19 | 42 | 44 | 86 | 30 | 29 | 59
  T2: PMB2948 (B24) | 10.6 [6.2 to 18.0] | 6.9 [4.1 to 11.5] | 8.6 [6.1 to 12.2] | 6.0 [4.7 to 7.8] | 8.5 [6.4 to 11.3] | 7.2 [5.9 to 8.7] | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.3 [3.7 to 5.0] | 4.1 [3.9 to 4.4]
  T2: PMB2707 (B44): number analyzed (Participants) | 9 | 10 | 19 | 47 | 47 | 94 | 23 | 29 | 52
  T2: PMB2707 (B44) | 23.5 [9.3 to 59.4] | 21.1 [6.5 to 68.3] | 22.2 [11.2 to 43.9] | 22.1 [15.5 to 31.6] | 17.0 [11.8 to 24.4] | 19.4 [15.1 to 24.9] | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 40 [NA to NA] — CI was not estimable due to the lack of variability of geometric means.
  T3: PMB80 (A22): number analyzed (Participants) | 9 | 11 | 20 | 45 | 51 | 96 | 31 | 29 | 60
  T3: PMB80 (A22) | 80.6 [30.9 to 210.7] | 82.3 [36.5 to 185.8] | 81.6 [46.6 to 142.8] | 63.0 [44.5 to 89.3] | 71.4 [52.7 to 96.6] | 67.3 [53.7 to 84.3] | 8.6 [7.5 to 9.8] | 8.6 [7.7 to 9.6] | 8.6 [7.9 to 9.3]
  T3: PMB2001 (A56): number analyzed (Participants) | 9 | 10 | 19 | 47 | 48 | 95 | 24 | 30 | 54
  T3: PMB2001 (A56) | 109.7 [70.4 to 171.1] | 181.0 [68.6 to 477.9] | 142.8 [85.5 to 238.6] | 190.6 [146.9 to 247.4] | 154.4 [116.3 to 205.1] | 171.4 [141.6 to 207.4] | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.3 [3.7 to 4.9] | 4.2 [3.8 to 4.5]
  T3: PMB2948 (B24): number analyzed (Participants) | 9 | 11 | 20 | 45 | 50 | 95 | 31 | 29 | 60
  T3: PMB2948 (B24) | 20.2 [11.1 to 36.6] | 17.0 [8.2 to 35.5] | 18.4 [11.8 to 28.6] | 15.8 [11.4 to 21.8] | 14.5 [11.1 to 19.1] | 15.1 [12.3 to 18.6] | 4.3 [3.7 to 4.9] | 4.4 [3.8 to 5.0] | 4.3 [3.9 to 4.8]
  T3: PMB2707 (B44): number analyzed (Participants) | 9 | 10 | 19 | 47 | 47 | 94 | 24 | 30 | 54
  T3: PMB2707 (B44) | 29.6 [11.6 to 75.8] | 34.3 [15.0 to 78.2] | 32.0 [18.3 to 55.8] | 46.3 [31.6 to 67.8] | 44.9 [31.3 to 64.5] | 45.6 [35.2 to 59.0] | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means.
  T4: PMB80 (A22): number analyzed (Participants) | 10 | 10 | 20 | 46 | 51 | 97 | 30 | 28 | 58
  T4: PMB80 (A22) | 10.6 [6.5 to 17.0] | 8.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 9.2 [7.3 to 11.5] | 10.8 [8.7 to 13.5] | 9.0 [7.9 to 10.2] | 9.8 [8.7 to 11.1] | 8.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 8.8 [7.5 to 10.4] | 8.4 [7.8 to 9.0]
  T4: PMB2001 (A56): number analyzed (Participants) | 8 | 10 | 18 | 41 | 47 | 88 | 24 | 28 | 52
  T4: PMB2001 (A56) | 7.3 [3.3 to 16.1] | 27.9 [11.3 to 68.5] | 15.4 [8.1 to 29.3] | 13.7 [9.4 to 20.1] | 12.5 [8.7 to 17.9] | 13.0 [10.1 to 16.9] | 4.1 [3.9 to 4.4] | 4.6 [3.4 to 6.3] | 4.4 [3.7 to 5.2]
  T4: PMB2948 (B24): number analyzed (Participants) | 10 | 10 | 20 | 46 | 51 | 97 | 30 | 28 | 58
  T4: PMB2948 (B24) | 4.9 [3.5 to 6.9] | 4.6 [3.4 to 6.3] | 4.8 [3.9 to 5.9] | 4.4 [4.0 to 4.9] | 4.9 [4.2 to 5.8] | 4.7 [4.2 to 5.2] | 4.1 [3.9 to 4.3] | 4.3 [3.7 to 5.0] | 4.2 [3.9 to 4.5]
  T4: PMB2707 (B44): number analyzed (Participants) | 8 | 8 | 16 | 43 | 46 | 89 | 24 | 29 | 53
  T4: PMB2707 (B44) | 4.8 [3.2 to 7.2] | 8.7 [2.6 to 29.5] | 6.4 [3.6 to 11.5] | 7.9 [5.8 to 10.6] | 7.3 [5.7 to 9.3] | 7.6 [6.3 to 9.1] | 4.1 [3.9 to 4.4] | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.1 [3.9 to 4.2]
  T5: PMB80 (A22): number analyzed (Participants) | 10 | 11 | 21 | 45 | 50 | 95 | 27 | 28 | 55
  T5: PMB80 (A22) | 8.6 [7.3 to 10.0] | 9.7 [7.2 to 13.1] | 9.1 [7.8 to 10.7] | 8.9 [7.9 to 10.0] | 8.6 [7.8 to 9.5] | 8.7 [8.1 to 9.4] | 8.2 [7.8 to 8.7] | 8.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 8.1 [7.9 to 8.3]
  T5: PMB2001 (A56): number analyzed (Participants) | 9 | 7 | 16 | 45 | 48 | 93 | 23 | 30 | 53
  T5: PMB2001 (A56) | 8.6 [3.4 to 22.1] | 35.3 [11.3 to 110.1] | 16.0 [7.6 to 33.5] | 7.9 [5.8 to 10.7] | 8.1 [6.0 to 11.0] | 8.0 [6.5 to 9.9] | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 5.3 [3.8 to 7.3] | 4.7 [3.9 to 5.6]
  T5: PMB2948 (B24): number analyzed (Participants) | 10 | 11 | 21 | 44 | 49 | 93 | 27 | 28 | 55
  T5: PMB2948 (B24) | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 5.1 [3.5 to 7.5] | 4.6 [3.8 to 5.5] | 4.1 [3.9 to 4.2] | 4.4 [3.8 to 5.0] | 4.2 [3.9 to 4.5] | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.6 [3.7 to 5.8] | 4.3 [3.9 to 4.8]
  T5: PMB2707 (B44): number analyzed (Participants) | 9 | 7 | 16 | 43 | 47 | 90 | 22 | 29 | 51
  T5: PMB2707 (B44) | 4.3 [3.6 to 5.2] | 4.9 [3.0 to 7.9] | 4.6 [3.7 to 5.6] | 5.3 [4.4 to 6.6] | 5.0 [4.2 to 5.9] | 5.2 [4.5 to 5.9] | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.1 [3.9 to 4.3] | 4.1 [3.9 to 4.2]
  T6: PMB80 (A22): number analyzed (Participants) | 10 | 9 | 19 | 34 | 47 | 81 | 0 | 0 | 0
  T6: PMB80 (A22) | 8.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 8.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 8.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 8.9 [7.6 to 10.3] | 8.4 [7.6 to 9.1] | 8.6 [7.9 to 9.3] |  |  |
  T6: PMB2001 (A56): number analyzed (Participants) | 9 | 8 | 17 | 39 | 40 | 79 | 0 | 0 | 0
  T6: PMB2001 (A56) | 6.9 [2.0 to 23.8] | 16.0 [7.5 to 34.2] | 10.2 [5.1 to 20.6] | 5.1 [4.0 to 6.6] | 7.3 [5.1 to 10.5] | 6.1 [4.9 to 7.6] |  |  |
  T6: PMB2948 (B24): number analyzed (Participants) | 10 | 9 | 19 | 34 | 48 | 82 | 0 | 0 | 0
  T6: PMB2948 (B24) | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 5.4 [2.7 to 11.1] | 4.6 [3.4 to 6.3] | 4.9 [3.8 to 6.4] | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 4.4 [3.9 to 4.8] |  |  |
  T6: PMB2707 (B44): number analyzed (Participants) | 9 | 8 | 17 | 39 | 41 | 80 | 0 | 0 | 0
  T6: PMB2707 (B44) | 4.0 [NA to NA] — CI was not estimable due to the lack of variability of geometric means. | 5.2 [3.4 to 8.0] | 4.5 [3.7 to 5.5] | 4.8 [4.0 to 5.7] | 5.0 [4.0 to 6.3] | 4.9 [4.2 to 5.6] |  |  |

19. Secondary Outcome: Percentage of Participants Reporting Pre-specified Local Reactions Within 7 Days After Booster Vaccination
Description: Local reactions included pain at injection site, swelling and redness collected by using an e-diary. Pain at injection site was graded as: mild (does not interfere with activity), moderate (interferes with activity) and severe (prevents daily activity). A caliper was used to measure the redness or swelling area. Caliper units were converted to centimeters (cm) according to 1 caliper unit = 0.5 cm. Redness and swelling were graded as: none (0 cm) mild (0.5-2.0 cm), moderate (>=2.0 to 7.0 cm) and severe (>7.0 cm).
Time Frame: Within 7 days after booster vaccination
Population: Booster safety population included all participants who received the booster dose at 23 months after vaccination 3 (Visit 12), and for whom safety information was available.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 120-mcg Bivalent rLP2086: Stage 2 Booster Phase: Participants who were randomly assigned to bivalent rLP2086 (irrespective of dose level) were eligible for booster vaccination. Participants received intramuscular injection of 120-mcg of bivalent rLP2086 vaccine after 23 months of visit 3.
Arm/Group | 120-mcg Bivalent rLP2086: Stage 2 Booster Phase
Number analyzed (Participants) | 147
percentage of participants
  Pain at injection site: mild | 30.6 [23.3 to 38.7]
  Pain at injection site: moderate | 29.3 [22.0 to 37.3]
  Pain at injection site: severe | 10.2 [5.8 to 16.3]
  Redness: mild | 22.4 [16.0 to 30.1]
  Redness: moderate | 21.1 [14.8 to 28.6]
  Redness: severe | 4.8 [1.9 to 9.6]
  Swelling: mild | 18.4 [12.5 to 25.6]
  Swelling: moderate | 15.0 [9.6 to 21.8]
  Swelling: severe | 0.0 [0.0 to 2.5]

20. Secondary Outcome: Percentage of Participants Reporting Systemic Events and Antipyretic Use Within 7 Days After Booster Vaccination
Description: Systemic reactions included fever, vomiting, diarrhea, headache, fatigue, muscle pain and joint pain were recorded by using an e-diary. Fever was defined as a temperature of greater than or equal to (>=) 38.0 degree Celsius and was graded as 38.0 degree Celsius (C) to 38.4 degree C, 38.5 degree C to 38.9 degree C, 39.0 degree C to 39.4 degree C, 39.5 degree C to 40.0 degree C, >40.0 degree C. Vomiting was graded as mild (1 to 2 times in 24 hours), moderate (>2 times in 24 hours) and severe (requires IV hydration). Diarrhea was graded as mild (2 to 3 loose stools in 24 hours), moderate (4 to 5 loose stools in 24 hours), and severe (6 or more loose stools in 24 hours). Fatigue, headache, muscle pain and joint pain were graded as: mild (did not interfere with activity), moderate (some interference with activity) and severe (prevented daily routine activity). The use and type of antipyretic medication was also recorded in the e-diary daily.
Time Frame: Within 7 days after booster vaccination
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 120-mcg Bivalent rLP2086: Stage 2 Booster Phase
Number analyzed (Participants) | 147
percentage of participants
  Fever >=38 degree C | 10.2 [5.8 to 16.3]
  Fever 38 to <38.5 degree C | 6.1 [2.8 to 11.3]
  Fever 38.5 to <39 degree C | 3.4 [1.1 to 7.8]
  Fever 39 to <39.5 degree C | 0.7 [0.0 to 3.7]
  Fever 39.5 to <=40 degree C | 0.0 [0.0 to 2.5]
  Fever >40 degree C | 0.0 [0.0 to 2.5]
  Vomiting: mild | 4.8 [1.9 to 9.6]
  Vomiting: moderate | 1.4 [0.2 to 4.8]
  Vomiting: severe | 0.0 [0.0 to 2.5]
  Diarrhea: mild | 4.8 [1.9 to 9.6]
  Diarrhea: moderate | 0.7 [0.0 to 3.7]
  Diarrhea: severe | 0.0 [0.0 to 2.5]
  Headache: mild | 7.5 [3.8 to 13.0]
  Headache: moderate | 10.2 [5.8 to 16.3]
  Headache: severe | 1.4 [0.2 to 4.8]
  Fatigue: mild | 17.0 [11.3 to 24.1]
  Fatigue: moderate | 22.4 [16.0 to 30.1]
  Fatigue: severe | 6.8 [3.3 to 12.2]
  Muscle pain : mild | 6.1 [2.8 to 11.3]
  Muscle pain : moderate | 8.2 [4.3 to 13.8]
  Muscle pain : severe | 2.0 [0.4 to 5.4]
  Joint pain: mild | 4.1 [1.5 to 8.7]
  Joint pain: moderate | 6.1 [2.8 to 11.3]
  Joint pain: severe | 0.0 [0.0 to 2.5]
  Antipyretic medication use | 34.7 [27.0 to 43.0]

21. Secondary Outcome: Percentage of Participants With SAE, MAE, NDCMC From Booster Vaccination to 1 Month After Booster Vaccination, 1 Month After Booster Vaccination to 6 Months After Booster Vaccination and Booster Vaccination Through 6 Months After Booster Vaccination
Description: SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; lack of efficacy in an approved indication; important medical event. A MAE was defined as a non-serious AE that resulted in an evaluation at a medical facility. An NDCMC was defined as a disease or medical condition that was not identified prior to study start and was expected to be persistent or otherwise long-lasting in its effects.
Time Frame: Booster vaccination to 1 month after booster vaccination (T1), 1 month after booster vaccination to 6 months after booster vaccination (T2) and booster vaccination through 6 months after booster vaccination (T3)
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 120-mcg Bivalent rLP2086: Stage 2 Booster Phase
Number analyzed (Participants) | 147
percentage of participants
  SAE: T1 | 0.7 [0.0 to 3.7]
  SAE: T2 | 0.7 [0.0 to 3.7]
  SAE: T3 | 1.4 [0.2 to 4.8]
  MAE: T1 | 4.8 [1.9 to 9.6]
  MAE: T2 | 2.7 [0.7 to 6.8]
  MAE: T3 | 7.5 [3.8 to 13.0]
  NDCMC: T1 | 0.0 [0.0 to 2.5]
  NDCMC: T2 | 0.0 [0.0 to 2.5]
  NDCMC: T3 | 0.0 [0.0 to 2.5]

22. Secondary Outcome: Percentage of Participants With at Least 1 Adverse Event (AE) From Booster Vaccination to 1 Month After Booster Vaccination
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship.
Time Frame: Booster vaccination up to 1 month after booster vaccination
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 120-mcg Bivalent rLP2086: Stage 2 Booster Phase
Number analyzed (Participants) | 147
percentage of participants | 13.6 [8.5 to 20.2]

23. Secondary Outcome: Percentage of Participants With Immediate Adverse Event (IAE) After Booster Vaccination
Description: Immediate AE was defined as AEs occurring within the first 30 minutes after investigational product administration.
Time Frame: Within 30 minutes after booster vaccination
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 120-mcg Bivalent rLP2086: Stage 2 Booster Phase
Number analyzed (Participants) | 147
percentage of participants | 0.0 [0.0 to 2.5]

24. Secondary Outcome: Percentage of Participants With hSBA Titer >=LLOQ >=1:4, >=1:8, >=1:16, >=1:32, >=1:64 and >=1:128 for Each of the 4 Primary Test Strains Before Booster Vaccination, and 1 Month After Booster Vaccination
Description: Percentage of participants achieving hSBA titer >= LLOQ were computed along with corresponding 2-sided 95 % CIs. The LLOQ was 1:16 for A22 and 1:8 for A56, B24, and B44.
Time Frame: Before booster vaccination and 1 month after booster vaccination
Population: Booster evaluable immunogenicity population: participants eligible for study, randomized to 120 mcg bivalent rLP2086 during stage 1, received scheduled investigational products, had blood drawn prior to booster vaccination dose and post-booster vaccination blood drawn (Visit 13) within 28-42 days from booster vaccination (Visit 12) and had no important protocol deviation. N=number of participants evaluable for this outcome measure and number analyzed=participants evaluable at specific rows.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 120-mcg Bivalent rLP2086: Stage 2 Booster Phase
Number analyzed (Participants) | 69
percentage of participants
  PMB80 (A22): before booster vaccination | 2.9 [0.4 to 10.1]
  PMB80 (A22):1 month after booster vaccination: number analyzed (Participants) | 68
  PMB80 (A22):1 month after booster vaccination | 92.6 [83.7 to 97.6]
  PMB2001 (A56):before booster vaccination: number analyzed (Participants) | 66
  PMB2001 (A56):before booster vaccination | 15.2 [7.5 to 26.1]
  PMB2001 (A56):1 month after booster vaccination: number analyzed (Participants) | 68
  PMB2001 (A56):1 month after booster vaccination | 100.0 [94.7 to 100.0]
  PMB2948 (B24): before booster vaccination | 7.2 [2.4 to 16.1]
  PMB2948 (B24):1 month after booster vaccination | 92.8 [83.9 to 97.6]
  PMB2707 (B44): before booster vaccination: number analyzed (Participants) | 67
  PMB2707 (B44): before booster vaccination | 9.0 [3.4 to 18.5]
  PMB2707 (B44): 1 month after booster vaccination | 95.7 [87.8 to 99.1]

25. Secondary Outcome: Serum Bactericidal Assay Using Human Complement (hSBA) Geometric Mean Titers (GMTs) for Each of the 4 MnB Primary Test Strains at Before Booster Vaccination and 1 Month After Booster Vaccination
Description: The LLOQ was 1:16 for A22, 1:8 for A56, B24, and B44. Titers below the LLOQ were set to 0.5*LLOQ for analysis. Titers were expressed in terms of 1/dilution.
Time Frame: Before booster vaccination and 1 month after booster vaccination
Population: as for outcome 24
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 120-mcg Bivalent rLP2086: Stage 2 Booster Phase
Number analyzed (Participants) | 69
titer
  PMB80 (A22): before booster vaccination | 8.4 [7.8 to 9.0]
  PMB80 (A22):1 month after booster vaccination: number analyzed (Participants) | 68
  PMB80 (A22):1 month after booster vaccination | 112.1 [87.2 to 144.2]
  PMB2001 (A56):before booster vaccination: number analyzed (Participants) | 66
  PMB2001 (A56):before booster vaccination | 5.2 [4.4 to 6.2]
  PMB2001 (A56):1 month after booster vaccination: number analyzed (Participants) | 68
  PMB2001 (A56):1 month after booster vaccination | 248.3 [192.7 to 319.9]
  PMB2948 (B24): before booster vaccination | 4.5 [4.0 to 5.1]
  PMB2948 (B24):1 month after booster vaccination | 48.3 [37.6 to 62.0]
  PMB2707 (B44): before booster vaccination: number analyzed (Participants) | 67
  PMB2707 (B44): before booster vaccination | 4.4 [4.1 to 4.9]
  PMB2707 (B44): 1 month after booster vaccination | 98.6 [71.4 to 136.2]

ADVERSE EVENTS:
Time Frame: Stage 1: SAEs:Recorded from Vaccination(Vacc) 1 through 6 months after Vacc. 3 (Month 12). Local reactions and systemic events in e-diary: 7 days after Vacc 1, 2 and 3. NSAEs: Vaccination 1 through 1 month after Vacc 3 (Month 7). Stage 2 Follow up phase: Month 24 visit (up to 30 days). Stage 2 Booster phase: SAEs: From booster vacc up to 6 months after booster vacc NSAEs: From booster vacc up to 1 month after booster vacc. Local reactions and systemic events in e-diary: 7 days after booster vacc
Description: SAEs and AEs were grouped by system organ class and preferred term. AEs included AEs collected in the e-diary (local and systemic reactions; systematic assessment) and AEs collected on the case report form at each visit (nonsystematic assessment).
Groups:
- Group 1: 60- Microgram (mcg) Bivalent rLP2086 (>=12 Months to <24 Months): Stage 1: Participants from greater than or equal to (>=) 12 months to less than (<) 24 months of age, received intramuscular injection of 60 mcg of bivalent rLP2086 vaccine on months 0 (visit 1, vaccination1), 2 (visit 4, vaccination 2), and 6 (visit 6, vaccination 3).
- Group 2: 120-mcg Bivalent rLP2086 (>=12 Months to <24 Months):Stage 1: Participants from >=12 months to <24 months of age, received intramuscular injection of 120 mcg of bivalent rLP2086 vaccine on months 0 (visit 1, vaccination1), 2 (visit 4, vaccination 2), and 6 (visit 6, vaccination 3). All eligible participants (who received 3 doses of bivalent rLP2086 in stage 1 at the 120 mcg dose level) received intramuscular injection of single booster dose of 120 mcg of bivalent rLP2086 after 23 months of vaccination 3 (visit 12) in stage 2. Participants were followed up approximately 6 months after the booster vaccination.
- Group 1: 60-mcg Bivalent rLP2086 (>=12 Months to <24 Months): Follow up: Participants from >=12 months to <24 months of age, received intramuscular injection of 60 µg of bivalent rLP2086 vaccine on months 0 (visit 1, vaccination1), 2 (visit 4, vaccination 2), and 6 (visit 6, vaccination 3).
- Group 2: 120-mcg Bivalent rLP2086 (>=12 Months to <24 Months): Follow up: Participants from >=12 months to <24 months of age, received intramuscular injection of 120 µg of bivalent rLP2086 vaccine on months 0 (visit 1, vaccination1), 2 (visit 4, vaccination 2), and 6 (visit 6, vaccination 3).
- Group 3: HAV/Saline (>=12 Months to <24 Months): Follow up: Participants from >=12 months to <24 months of age, received intramuscular injection of saline on 2- month and HAV vaccine on months 0 (visit 1, vaccination1), 2 (visit 4, vaccination 2), and 6 (visit 6, vaccination 3).
Arm/Group | Group 1: 60- Microgram (mcg) Bivalent rLP2086 (>=12 Months to <24 Months): Stage 1 | Group 2: 120-mcg Bivalent rLP2086 (>=12 Months to <24 Months):Stage 1 | Group 3: HAV/Saline (>=12 Months to <24 Months): Stage 1 | 120-mcg Bivalent rLP2086: Stage 2 Booster Phase | Group 1: 60-mcg Bivalent rLP2086 (>=12 Months to <24 Months): Follow up | Group 2: 120-mcg Bivalent rLP2086 (>=12 Months to <24 Months): Follow up | Group 3: HAV/Saline (>=12 Months to <24 Months): Follow up
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/220 | 0/132 | 0/147 | 0/44 | 0/220 | 0/132
Serious Adverse Events (participants affected / at risk) | 4/44 | 19/220 | 8/132 | 2/147 | 0/44 | 3/220 | 0/132
Other Adverse Events (participants affected / at risk) | 43/44 | 209/220 | 113/132 | 121/147 | 0/44 | 0/220 | 0/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: 60- Microgram (mcg) Bivalent rLP2086 (>=12 Months to <24 Months): Stage 1 (N=44) | Group 2: 120-mcg Bivalent rLP2086 (>=12 Months to <24 Months):Stage 1 (N=220) | Group 3: HAV/Saline (>=12 Months to <24 Months): Stage 1 (N=132) | 120-mcg Bivalent rLP2086: Stage 2 Booster Phase (N=147) | Group 1: 60-mcg Bivalent rLP2086 (>=12 Months to <24 Months): Follow up (N=44) | Group 2: 120-mcg Bivalent rLP2086 (>=12 Months to <24 Months): Follow up (N=220) | Group 3: HAV/Saline (>=12 Months to <24 Months): Follow up (N=132)
Eyelid ptosis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Crying (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Bronchiolitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Bronchitis (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Croup infectious (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Enterovirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Gastroenteritis (Infections and infestations) | 0 | 3 | 1 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Otitis media (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Otitis media chronic (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Pneumonia (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Tonsillitis (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Viral tonsillitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Balance disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Cerebellar ataxia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Irritability (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Polydipsia psychogenic (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Rhinovirus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: 60- Microgram (mcg) Bivalent rLP2086 (>=12 Months to <24 Months): Stage 1 (N=44) | Group 2: 120-mcg Bivalent rLP2086 (>=12 Months to <24 Months):Stage 1 (N=220) | Group 3: HAV/Saline (>=12 Months to <24 Months): Stage 1 (N=132) | 120-mcg Bivalent rLP2086: Stage 2 Booster Phase (N=147) | Group 1: 60-mcg Bivalent rLP2086 (>=12 Months to <24 Months): Follow up (N=44) | Group 2: 120-mcg Bivalent rLP2086 (>=12 Months to <24 Months): Follow up (N=220) | Group 3: HAV/Saline (>=12 Months to <24 Months): Follow up (N=132)
Eustachian tube disorder (Ear and labyrinth disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Middle ear effusion (Ear and labyrinth disorders) | 0 | 8 | 3 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Anisometropia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Astigmatism (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Hypermetropia (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Aphthous ulcer (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Diarrhoea (Gastrointestinal disorders) | 1 | 11 | 5 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Teething (Gastrointestinal disorders) | 0 | 8 | 4 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Vomiting (Gastrointestinal disorders) | 1 | 8 | 5 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Chills (General disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Injection site erythema (redness) (General disorders) | 30 | 137 | 28 | 71 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Injection site erythema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Injection site pain (tenderness at injection site) (General disorders) | 35 | 160 | 41 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Injection site pain (General disorders) | 1 | 4 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Injection site swelling (swelling) (General disorders) | 17 | 103 | 20 | 49 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Pyrexia (fever) (General disorders) | 16 | 82 | 20 | 15 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Pyrexia (General disorders) | 1 | 18 | 6 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Vaccination site pain (General disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Vessel puncture site bruise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Food allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Bronchiolitis (Infections and infestations) | 0 | 3 | 2 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Bronchitis (Infections and infestations) | 5 | 22 | 11 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Cellulitis (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Conjunctivitis (Infections and infestations) | 1 | 22 | 13 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Croup infectious (Infections and infestations) | 0 | 9 | 2 | 2 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Enterobiasis (Infections and infestations) | 0 | 2 | 2 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Exanthema subitum (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Gastroenteritis viral (Infections and infestations) | 1 | 10 | 3 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Gastroenteritis (Infections and infestations) | 4 | 29 | 11 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Hand-foot-and-mouth disease (Infections and infestations) | 2 | 10 | 6 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Impetigo (Infections and infestations) | 1 | 3 | 3 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Infected bite (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Laryngitis (Infections and infestations) | 2 | 3 | 5 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Lower respiratory tract infection (Infections and infestations) | 0 | 4 | 2 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Molluscum contagiosum (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Nasopharyngitis (Infections and infestations) | 7 | 3 | 7 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Otitis externa (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Otitis media acute (Infections and infestations) | 1 | 2 | 2 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Otitis media (Infections and infestations) | 3 | 27 | 20 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Pharyngitis (Infections and infestations) | 6 | 18 | 15 | 2 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Pharyngotonsillitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Pneumonia (Infections and infestations) | 0 | 7 | 2 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Respiratory tract infection viral (Infections and infestations) | 2 | 3 | 1 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Respiratory tract infection (Infections and infestations) | 0 | 4 | 1 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Rhinitis (Infections and infestations) | 3 | 8 | 3 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Skin candida (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Tonsillitis (Infections and infestations) | 4 | 6 | 9 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Tracheitis (Infections and infestations) | 1 | 1 | 5 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Upper respiratory tract infection (Infections and infestations) | 6 | 58 | 34 | 3 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Urinary tract infection (Infections and infestations) | 0 | 7 | 3 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Varicella (Infections and infestations) | 2 | 5 | 3 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Viral infection (Infections and infestations) | 1 | 3 | 2 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Viral pharyngitis (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Viral tonsillitis (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Viral upper respiratory tract infection (Infections and infestations) | 5 | 45 | 23 | 5 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 3 | 1 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Contusion (Injury, poisoning and procedural complications) | 0 | 5 | 2 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Fall (Injury, poisoning and procedural complications) | 2 | 5 | 7 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Laceration (Injury, poisoning and procedural complications) | 1 | 4 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Lip injury (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Decreased appetite (loss of appetite) (Metabolism and nutrition disorders) | 22 | 142 | 50 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 2 | 2 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Somnolence (drowsiness) (Nervous system disorders) | 23 | 127 | 40 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Somnolence (Nervous system disorders) | 0 | 3 | 2 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Irritability (Psychiatric disorders) | 5 | 21 | 5 | 2 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 8 | 3 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 11 | 2 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 4 | 2 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 4 | 1 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Eczema (Skin and subcutaneous tissue disorders) | 0 | 4 | 4 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Miliaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 4 | 2 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Irritability (Psychiatric disorders) | 31 | 176 | 69 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 3 | 3 | 0 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 9 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Fatigue (General disorders) | 0 | 0 | 0 | 68 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Injection site pain (General disorders) | 0 | 0 | 0 | 103 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 15 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 24 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Headache (Nervous system disorders) | 0 | 0 | 0 | 28 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups.
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 8 | 0 | 0 | 0 — MedDRA v20.0 for Group 1: 60mcg bivalent rLP2086 (>=12 months to <24 months), Group 2: 120mcg bivalent rLP2086 (>=12 months to <24 months), Group 3: HAV/Saline (>=12 months to <24 months); MedDRA v23.0 for booster stage and safety follow up groups

LIMITATIONS AND CAVEATS:
The immunogenicity data at 36 and 48 months after vaccination 3 was not collected due to change in planned analysis as per latest protocol amendment, according to which blood draw of participants at 36 and 48 months after Vaccination 3 was removed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-04-19): https://cdn.clinicaltrials.gov/large-docs/35/NCT02534935/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-13): https://cdn.clinicaltrials.gov/large-docs/35/NCT02534935/SAP_001.pdf